

## INSTITUTIONAL REVIEW BOARD RECOMMENDATION

#### CONTINUING REVIEW

Date of Review:

30 May 2018

Protocol Number: NHRC.2016.0019

Protocol Title:

Evaluation of a Mobile Application for Prescription Drug-Abuse Education (MAPDE)

Principal Investigator:

Suzanne Hurtado, MPH

Work Unit title/#/JON:

Mobile Tools for Risk Reduction and Health Promotion for Military Members,

N1514; JON: 8ZE123

The principal investigator submitted a continuing review application for a protocol that was previously classified as minimal risk. The purpose of this study is to test a new smartphone application ("app") called MAPDE, to educate about prescription drug abuse. This app was built to help military members reduce their risk of prescription drug misuse. The app contains various educational sections and tools such as: selfassessments for risk of misuse with tailored feedback and recommendations; information on misuse, drug interactions and more; scenarios to practice communication skills related to preventing misuse; resources for help and more. About 60 to 80 active-duty Navy or Marine Corps military members, 18 years or older, will be invited to participate in this study. Consenting participants will complete an online survey about prescription drug use, knowledge and attitudes related to prescription drug misuse, and mental well-being. Participants will be randomly assigned to one of two groups: 1) use the smartphone app for this study and continue with their physician's care and treatment as usual; or 2) continue with their physician's care and treatment as usual without the smartphone app. No names or personally identifiable information will be collected for this study. This effort has been requested and funded by the National Institute on Drug Abuse. A Cooperative Research and Development Agreement (CRADA; NHRC-14-9374) with Intelligent Automation, Inc. is currently in place. Survey approval has been obtained from OPNAV (OPNAV RCS 6320-5) and USMC (USMC-IR-17002). To date, 81 subjects have been studied. Subject enrollment is complete. The principal investigator indicated that there have been no untoward events, complications, or injuries.

The continuing review requests to 1) add Stephanie Kewley (Leidos) as key support personnel to the protocol and 2) remove Kyle O'Donnell. The principal investigator indicated compliance with all relevant human subject protection regulations.

The Chair reviewed this continuing review under the expedited review authority permitted under 32 CFR § 219.11 (b)(2). The criteria for the approval of research continue to be met under 32 CFR § 219.111. The NHRC Chair recommends approval of this research.

The current IRB approval period expires on 14 June 2019.

W.J. BECKER, Ph.D. Chair, NHRC IRB

WJ/Secher Signature

05/31/20/8



# DETERMINATION OF APPROVING AUTHORITY

| 1.) | I concur with the recommendation of the IRB, and I approve continuation of this research. |
|---|---|
| | FF |

Next review is required no later than: 14 June 2019

I concur with the recommendations of the IRB, but I require additional modifications or restrictions prior to providing continuing approval (Attach modifications or restrictions required).

Next review is required no later than:

3. I disagree with the recommendations of the IRB and recommend (Attach statement regarding recommendations and reasons).

Signature

Date (MM/DD/YY)

M. R. MONTEVILLE, CAPT, MSC, USN Commanding Officer

MITT

06/04/18

| HUMAN USE PROTOCOL<br>ROUTING SLIP | | | | | | |
|---|---|---|---|---|---|---|
| Suza | M (Principal Investigator):<br>nne L. Hurtado, MPH<br>PED NAME) | Sezame Horszlo-<br>(PI SIGNATURE) | | | | |
| | In accordance with NAVHLTHRSCHCENINST 3900.2G, I am submitting the attached human use protocol for consideration. | | | | | |
| TITL | E OF PROTOCOL: Evaluation | n of a Mobile A | pplication fo | r Prescripti | on Drug Abuse | Education |
| ABB | ABBREVIATED TITLE: Evaluation of a Drug Abuse Educational App | | | | | |
| PRO | POSED DATES OF RESEARC | CH: 2016JUN0 | 1 to 2019JUN | V01 | | |
| FUN | DING SOURCE: National Inst | itute on Drug A | buse via Inte | lligent Aut | omation Inc. (p | rimary awardee) |
| WOR<br>N151 | K UNIT TITLE AND NUMB<br>4 | ER: Mobile Too | ls for Risk R | eduction a | nd Health Prom | notion for Military Members, |
| JON | FUNDING THE PROTOCOL: | 8ZE123 | | | | |
| SUB | MISSION (CHECK ONE): | | | | | |
| ☐ INITIAL SUBMISSION ☐ MODIFICATION OF PREVIOUS SUBMISSION ☑ CONTINUING/ANNUAL REVIEW | | | | | | |
| | TOCOL OBJECTIVE (Brief se | | | | | application for prescription |
| drug abuse education to determine feasibility and potential for effectiveness. | | | | | | |
| DoD PROTOCOL NUMBER (Assigned by IRB Administrator upon submission for initial review. Be sure to add this | | | | | | |
| number where indicated on the title page): NHRC.2016.0019 | | | | | | |
| signa | You must obtain required tures before you submit the col to the IRB. | Date<br>Received | Date<br>Reviewed | Initials | Approved<br>JON<br>Initials | NOTES |
| 1 | DEPARTMENT HEAD | 14 May 18 | | Cja | Cft | |
| 2 | DIRECTOR* | | | , | N/A | |
| 3 | CHIEF SCIENCE EXEC* | 4 1 0040 | | | N/A | |
| 4 | IRB ADMINISTRATOR | MAY 14 2018 | N/A | As C | N/A | |

From: Suzanne Hurtado

To: Chair, Institutional Review Board, Naval Health Research Center, San Diego, CA

Subj: CONTINUING REVIEW OF PROTOCOL #NHRC.2016.0019, Evaluation of a Mobile Application for Prescription Drug Abuse Education

Ref: (a) NAVHLTHRSCHCENINST 3900.2G

Encl: (1) Continuing Review Summary for Protocol #NHRC.2016.0019

(2) All subject materials for re-approval including recruitment materials, informed consent form, privacy act, surveys, etc. [If subject enrollment is ongoing] (N/A – subject enrollment is complete)

- (3) List of all current Study Personnel (with company affiliations and research role)
- (4) Full Current Protocol (clean and tracked-changes)
- (5) If applicable, Sponsor Protocol and Drug/Device Information (N/A)
- 1. Enclosure (1) is submitted to fulfill the reference (a) requirement for the Institutional Review Board (IRB) to review all work conducted under previously approved research protocols at least annually.
- 2. Point of contact for further information is Suzanne Hurtado at (619) 553-7806 or email: Suzanne.l.hurtado.civ@mail.mil.
- 3. I certify that all study personnel have been informed of and accept any proposed changes.

Suzanne Hurtado 14 May 2018

PI Signature and Date

#### CONTINUING REVIEW FOR IRB PROTOCOL NUMBER NHRC.2016.0019

- 1. PROTOCOL NUMBER: NHRC.2016.0019
- 2. <u>PROTOCOL TITLE</u>: Evaluation of a Mobile Application for Prescription Drug Abuse Education
- 3. <u>WORK UNIT TITLE AND NUMBER</u>: Mobile Tools for Risk Reduction and Health Promotion for Military Members, N1514
- 4. PRINCIPAL INVESTIGATOR(S): Suzanne Hurtado, MPH

#### 5. <u>UPDATE OF RESEARCH BACKGROUND</u>

The research literature relevant to this project appearing in print since the last IRB review of this protocol has been surveyed. The research issues addressed in this research protocol have not been resolved. No additional risks or benefits have been identified from the review of the recent literature. Based on this review, the utility of the research and the risk-benefit ratio have not changed.

#### 6. CHANGES SINCE LAST REVIEW

- We request to extend the proposed dates of research to 2019JUN01 to allow another year for completion of analysis and manuscripts.
- We request to remove Kyle O'Donnell from the protocol as he has left NHRC.
- We request to add Stephanie Kewley to the protocol..

#### 7. SUBJECTS

The targeted sample size of this study was 60 to 80 participants. We have studied 81 subjects, all of whom were enrolled in the study. The circumstances that led to the study exceeding the maximum number of participants are that in the final days of the enrollment phase, there were several potential participants who had been consented and were invited to participate in the online survey. The 80<sup>th</sup> and 81<sup>st</sup> participants both formalized their consent and participated in the online survey after working hours (in the night time), so the PI did not have the opportunity to close enrollment right after the 80<sup>th</sup> participant. Since the 81<sup>st</sup> participant had begun their study participation and had been told they would receive the study incentive, we included them. Subject enrollment is complete.

#### 8. ADVERSE/UNEXPECTED EVENTS

There have been no untoward events, complications, or injuries.

## 9. MEDICAL CARE

It has not been necessary to provide medical care to any study participants.

#### 10. INFORMED CONSENT

Informed consent has been obtained from all study participants by providing them with a PDF copy of the consent form approved by the IRB, and participants should have read the consent form on the study website as well. They were given time to read it, and they were encouraged to contact the PI with any questions they may have had about the protocol at any time. The voluntary nature of participation was

stressed, and no supervisors or superior officers who might have applied pressure to coerce participation were involved in the process. Per the approved IRB protocol, consent to participant was obtained using a web-based consent form, in which the participant clicked the appropriate box ("I consent" or "I do NOT consent").

#### 11. RESEARCH AND SAFETY PROCEDURES

All research and safety procedures have faithfully conformed to the descriptions in the protocol as approved by the IRB.

#### 12. FINDINGS TO DATE

Follow-up data collection is still in progress. There are no research findings to report at this time.

#### 13. <u>COMPLIANCE WITH REGULATIONS</u>

To the best of my knowledge, this project has been conducted in compliance with all of the requirements of NAVHLTHRSCHCENINST 3900.2G and the related instructions and regulations cited therein.

#### 14. PERSONNEL QUALIFICATIONS

All personnel are appropriately trained and qualified for their work on the project.

#### 15. MAINTENANCE OF RECORDS

All IRB-relevant records are properly kept and securely stored as described in the protocol approved by the IRB.

#### 16. CONFLICT OF INTEREST

No persons involved in the design, conduct, or reporting of research has a financial or other interest that could reasonably appear to be affected by the carrying out or the results of the research.

#### 17. COLLABORATING INSTITUTIONS

This protocol does not involve collaboration with any other institutions, so there has not been and will not be a continuing review by any other Institutional Review Board.

PI Signature and Date

| HUMAN USE PROTOCOL<br>ROUTING SLIP – INITIAL SUBMISSION | | | | |
|---|---|---|---|---|
| Suza | M (Principal Investigator):<br>nne Hurtado, MPH<br>PED NAME) | | | |
| | | (PI SIGNATURE) | | |
| | In accordance with NAVHLTHRSCHCENINST 3900.2G, I am submitting the attached human use protocol for consideration. | | | |
| TITI | E OF PROTOCOL: Evaluation of a M | obile Application for Pres | scription Drug Abuse Edu | ucation |
| ABBREVIATED TITLE: Evaluation of a Drug Abuse Educational App | | | | |
| PRO | POSED DATES OF RESEARCH: 20 | 016MAY01 to 2018MAY | 01 | |
| FUN | DING SOURCE: National Institute on | Drug Abuse via Intelliger | nt Automation Inc. (prima | ary awardee) |
| WORK UNIT TITLE AND NUMBER: Mobile Tools for Risk Reduction and Health Promotion for Military Members, N1514 | | | | |
| LIFE OF FUNDING (number of years): 1 year with 1 additional option year | | | | |
| SUBMISSION (CHECK ONE): INITIAL SUBMISSION MODIFICATION OF PREVIOUS SUBMISSION CONTINUING/ANNUAL REVIEW | | | | |
| PROTOCOL OBJECTIVE (Brief sentence or two): Conduct a test of a smartphone mobile application for prescription drug abuse education to determine feasibility and potential for effectiveness. | | | | |
| DoD PROTOCOL NUMBER (Assigned by IRB Administrator upon submission for initial review. Be sure to add this number where indicated on the title page): NHRC.2016.0019 | | | | |
| repre | Note: You must obtain Dept. IRB representative signature before you submit the protocol to the IRB. DATE RECEIVED DATE APPROVED INITIALS | | | |
| 1 | DEPARTMENT IRB MEMBER | 8 | | |
| 2 | IRB ADMINISTRATOR | | | |

#### I. COVER PAGE(S)

1. Protocol Number:

NHRC.2016.0019

2. Title:

Evaluation of a Mobile Application for Prescription Drug Abuse Education

3. Date of Submission: 01 MAY 2016

4. Approved Work Unit Title (i.e., the funded research proposal [or also referred to as the work unit] title under which the protocol is being conducted) and Full Work Unit Number:

Mobile Tools for Risk Reduction and Health Promotion for Military Members, N1514

- Approximate Dates of Research (in yyyymmmdd format, e.g., 1996DEC12): 2016MAY01 to 2018MAY01
- Principal Investigator: Suzanne L. Hurtado, MPH Naval Health Research Center

7. Co-Investigator(s):

Cynthia M. Simon-Arndt

Leidos Inc. contractor, Naval Health Research Center

Cynthia J. Thomsen

Naval Health Research Center

8. Key Support:

Renee Dell'Acqua

Leidos contractor, Naval Health Research Center

Elizabeth Lauer

Leidos contractor, Naval Health Research Center

Robyn Martin

Leidos contractor, Naval Health Research Center

Shannon Fitzmaurice

Leidos contractor, Naval Health Research Center

Casey Kohen

Leidos contractor, Naval Health Research Center

Stephanie Kewley

Leidos contractor, Naval Health Research Center

9. Identification Research Monitor/Ombudsman: N/A

10. Primary Performing Institution(s):

Naval Health Research Center

11. Collaborating Institution(s):

N/A

i

12. Funding Source:

National Institute on Drug Abuse via CRADA with Intelligent

Automation, Inc.

13. Subjects:

a. Number of Subjects: 80

- b. Number of Female Subjects: 14
- c. Number of Male Subjects: 66
- d. Number of Civilian Subjects: 0
- e. Number of Active-Duty Subjects: 80
- 14. Is an IAIR/IIRR needed? No

# II. SIGNATURE PAGE

| 1. | Principal Investigator | Suzanne L. Hurtado, MPH Naval Health Research Center |
|---|---|---|
| 2. | Directorate Head/Dept. Head | Dennis Faix, MD, MPH/CDR, MC, USN<br>Head, Military Population Health Directorate/<br>Cynthia Thomsen, PhD, Department Head, Health and<br>Behavioral Sciences |
| 3. | Principal Director of Research | Richard Shaffer, PhD |
| 4. | Ombudsman (if applicable) | N/A |
| 5. | Research Monitor (if applicable) | N/A |
| 6. | Commanding Officer: | R. G. SIMMONS, CAPT, MSC, USN |

#### III. RECORD OF CHANGES TO THE PROTOCOL

5/14/2018 — A continuing review was submitted, which included a request to remove Kyle O'Donnell and to extend the research till 2019JUN01 to complete analyses and reports.

10/4/2017 - A modification was approved to replace Rosemarie Subala with Kyle O'Donnell.

9/13/2017 - A modification was approved to add Elizabeth Lauer, Robyn Martin, Shannon Fitzmaurice and Casey Kohen.

iv

5/15/2017 – A continuing review was approved that added Renee Dell'Acqua and removed Steven Hanling.

## IV. TABLE OF CONTENTS

| I. COVER PAGE(S) |
|---|
| II. SIGNATURE PAGE |
| III. RECORD OF CHANGES TO THE PROTOCOL |
| IV. TABLE OF CONTENTS |
| V. SCIENTIFIC BACKGROUND AND OBJECTIVES 1. Background 2. Objectives A. Hypothesis(es) to be tested B. Other objective(s) |
| VI. EXPERIMENTAL METHODS 1. Experimental Procedures and Rationale A. Subjects B. Methods and Informed Consent Plan 2. Sample Size Determination With Statistical Power Calculation 3. Justification for Exclusion of Specific Groups 4. Required Equipment and Supplies. |
| VII. ORGANIZATION OF RESEARCH EFFORT |
| VIII. RISKS AND DISCOMFORTS TO RESEARCH VOLUNTEERS |
| IX. DESCRIPTION OF THE SYSTEM FOR MAINTENANCE OF RECORD 1. Experimental Data |
| X. APPENDICES A. VOLUNTARY CONSENT TO PARTICIPATE IN A RESEARCH STUDY B. INVESTIGATOR COMPLIANCE ATTESTATION C. REFERENCES D. LIST OF MEDICATIONS E. FLYER F. SURVEY INVITATIONS AND REMINDERS F- |

#### V. SCIENTIFIC BACKGROUND AND OBJECTIVES

#### 1. Background

In a recent review of military substance abuse treatment and prevention, the Institute of Medicine concluded that substance use and misuse have reached the level of a public health crisis within the armed forces (O'Brien et al., 2012). Research regarding military substance use suggests that certain substance problems, particularly prescription drug misuse, have increased significantly among military personnel over the last decade (Bray et al., 2010). Furthermore, prescription drug misuse in the prior 30 days is higher among military personnel than similar civilians (12% vs. 4%; Bray, Pemberton, Hourani et al., 2009). Higher rates of prescription drug misuse in the military may be driven in part by dramatic increases in prescriptions for medications (including psychoactive and pain medications) issued to military members since the beginning of the OIF/OEF era (Friedman, 2013; Zoroya, 2010). In contrast, most likely due to strict zero tolerance policies, the prevalence of illicit drug use in the prior 30 days is remarkably low among military personnel relative to civilians 2% vs. 12% (Bray, Pemberton, Hourani et al., 2009). Expanded drug testing protocols that test for additional prescription compounds also reflect the higher levels of prescription drug misuse compared with other drugs, and measures to reduce the trend are deemed important to readiness by the Department of the Navy (DoN, 2015).

At the same time, the Department of Defense has invested heavily in smartphone app technology for use on military networks (http://www.defense.gov/news/newsarticle.aspx?id=120388), as well as through the DARPA Transformative Apps program. However, no existing application targets prescription drug misuse. Given the growing ownership and use of smartphones by military personnel, an evidence-based prescription drug-abuse prevention program delivered through a mobile application (app) would address an important gap in substance abuse prevention for military personnel.

To address this identified need, technology developers at Intelligent Automation, Inc. and researchers at the Naval Health Research Center have developed an evidence-based prescription drug-abuse prevention mobile app prototype called MAPDE (Mobile Application for Prescription Drug-Abuse Education). MAPDE will help military members reduce prescription drug misuse by enhancing critical communication and decision-making skills. Ideally, military members will use the program and modify high-risk behavior before addiction and serious negative consequences occur. This prevention and skills-building tool is intended to augment in-person medical visits and other educational programs, such as Prescription for Discharge, as one component of a multi-faceted effort to reduce prescription drug misuse among military members. This program will provide a way for service members to learn more about reducing prescription drug misuse and is a way of reaching members who may not want to access more formal resources due to stigma associated with substance abuse treatment.

Under a previous NHRC protocol (NHRC.2014.0042), the researchers conducted a usability test of the prototype app in collaboration with pain clinic physicians at Naval Medical Center San Diego. The test indicated positive findings about the usability of MAPDE; it received high scores on likability and appropriateness for a military population. In addition, some redesign issues were identified, which included improving the functionality of the My Meds section; improving the utility of the feedback on skipped questions in the Assessments module; and improving the usefulness and user satisfaction of the scenarios under the Practice module. These issues and other improvements are being addressed in a new version of the app, which will be tested. The current protocol describes the procedures for conducting a test of the app to evaluate feasibility and acceptability, and the potential impact of MAPDE on reducing misuse risks.

The effort has been requested and funded by the National Institute on Drug Abuse. Intelligent Automation, Inc. is the direct recipient of a Phase 2 small business development grant and is funding NHRC's contribution to the effort, which is to support content development and conduct a test of the mobile application.

#### 2. Objectives

A. Hypothesis(es) to be tested

(1) Participants receiving the mobile application plus treatment as usual will have lower

prescription drug misuse risk scores, greater knowledge and improved attitudes compared to participants receiving treatment as usual only.

- B. Other objective(s)
- (1) Assess the feasibility and acceptability of the mobile application.

#### VI. EXPERIMENTAL METHODS

#### 1. Experimental Procedures and Rationale

#### A. Subjects

Eighty active duty participants will be initially recruited for this study. Potential participants will be patients of the pain clinic, deployment health clinic and other primary care clinics, or pharmacy patrons of the Naval Medical Center San Diego (NMCSD) who have currently been prescribed a medication(s) with the potential for misuse. The participants will likely reflect the demographics of the overall Navy population. The percentage of women in the Navy is approximately 17% and the age range of the sample is expected to be 18 to 55 years of age. The sample is also expected to include a variety of racial groups and ranks.

The inclusionary criteria are that the participant must be age 18 or older, on active-duty status, in the Navy or Marine Corps, have a current prescription for a medication with the potential for misuse, and own a smartphone (all to be confirmed verbally with participants prior to consent). A list of prescription medications with the potential for misuse will be used for this medication criterion; see Appendix D. The list was developed based on information from the National Institute on Drug Abuse, Commonly Abused Drugs Charts-prescription drugs; the Drug Enforcement Agency; and consultations with Navy pain clinic physicians and a Navy pharmacist. No potential participants will be excluded based on rank or other demographics.

#### B. Methods and Informed Consent Plan

Study design. The study consists of a randomized controlled design with two groups. The control group will be provided with treatment as usual, and the experimental group will be provided with the MAPDE smartphone application in addition to treatment as usual. Repeated measures will be administered to all participants at baseline, 1 month, and 3 months. This study does not propose any modification or change to the physician's treatment plan, and the app is not considered a medical device under section 201(h) of the Federal Food, Drug, and Cosmetic Act (FD&C Act). Study results will also be used to determine estimates of intervention effect sizes to be used in a later effectiveness trial. In addition, the study will determine the feasibility and acceptability of the mobile app.

In general, treatment as usual for a patient who is currently taking a prescribed medication is characterized as being under the care of a physician and receiving the prescribed care and treatment by that physician or medical team according to the patient's specific needs. For a patient who is a participant in the NMCSD Pain Clinic's functional and restorative pain program and who is currently taking a prescribed medication, their treatment as usual involves being under the care of a physician as part of the facility's broader pain program, which encompasses other components such as additional medical management of pain, physical rehabilitation, and psychological therapy. Regardless, it should be clear that this study is not interfering in any way with the patient's usual treatment.

Recruitment. Participants will be recruited from patient waiting rooms and medical offices of the NMCSD such as the pain clinic, primary care clinics, deployment health clinic and pharmacy waiting areas using two approaches. The first approach is using flyers (see Appendix E) about the study opportunity that will be posted in the waiting areas, clinics and pharmacy. The flyer will

instruct potential participants to contact the Principal Investigator (PI) to learn more about the study. The second approach is an in-person approach to tell potential participants about the study opportunity. This will occur by having a research team member onsite in the pharmacy waiting room area handing out flyers and asking potential participants if they would be interested in the study. The in-person approach will also be used by the study's consultant who is also a provider in the pain clinic. When the provider sees a pain clinic patient, he will hand out a flyer and ask the potential participant if they would be interested in the study. In both cases, the staff member can explain more about the study, and go over the inclusionary criteria and answer any questions.

When the potential participant contacts the PI about the study, the PI will ask if the participant meets the inclusionary criteria. They will also emphasize that participation is voluntary. If they meet the criteria, the PI will then ask for their non-DoD email address to communicate with the participant during the study, and to link their surveys over time. Non-DoD email addresses are less likely to contain a person's full name compared to DoD email addresses. However, in the case that the potential participant is uncomfortable using their current non-DoD (personal) email address, we will provide instructions for setting up a new personal email account on Gmail if they would like to create a new email address for the study to further ensure their anonymity. The PI will send an email to the participant with the: (1) consent form in an attachment for their review; (2) a web link to access the survey website; and (3) instructions for creating a new personal email address for the study with a request to send that to the PI.

The PI or study staff will randomly assign the participant to a study condition, which will indicate which survey link or path, specific to the study condition that they will receive, and then the participant will be sent an email. Each email path will have identical consent documentation; however, this method enables the study team to tailor the follow up messaging more easily. The PI will maintain a list of participant emails and their study group assignment for the purpose of sending survey and intervention reminders.

Informed consent plan. The participant will have received a copy of the consent form in the email from the Pl. Also, once the participant accesses the web link (for either survey path—intervention group or control group), the first page they will see will be the consent page. If the participant has any questions, the form encourages the participant to contact the Pl and ask questions about the research. If the participant consents to participate, they will indicate this on the web-based consent form by clicking the appropriate box ("I consent" or "I do NOT consent"). If "I do NOT consent" is selected, a screen that thanks them for visiting the site will appear along with the standard instruction to close their browser. The participant must also check a box indicating that they attest that their participation is during off-duty, liberty or leave status. If the box is left unchecked by the participant, they may not be compensated for participating in the study.

**Procedures.** After the subject consents to participate, the website will also present them with a statement that requires the participant to agree, by checking a box, that their participation will only take place during their off-duty time. (The consent form also clearly instructs participants to complete the survey during their off-duty time.) Then they will be presented with the Privacy Act Statement.

The surveys will be web-based and the website will be hosted on a Qualtrics server that uses a high-end firewall system, transport layer security, passwords, and encryption. In order to deter individuals from taking the survey multiple times, Qualtrics' "Prevent Ballot Box Stuffing" feature will be used. This feature places a cookie on the respondent's browser, which will not allow them to use the survey link a second time.

Participants will be asked to enter their non-DoD email address as a way to link their surveys over time. Then, they will enter their responses online; their data will automatically be saved to a data file. Measures will be taken to protect the email addresses and survey data collected (see Risk to the Volunteer and Means of Mitigation, and Experimental Data sections).

After submitting the baseline survey, participants in the intervention group will get instructions for downloading the MAPDE app. They will be asked to download the app from the app store (e.g., iOS or Google app store), and they will be given a unique key number to access the app once downloaded. (The PI will log into the app developer's web portal for the app and manually create a unique key number that does not contain any PII information, and provide the key to the consenting participant.) The user will also be required to set up a separate self-selected 4-digit PIN and re-enter it each time they open the app, to further enhance security. Neither the participant's phone number nor any ID that can be used to identify the phone or its user will ever be stored in the app developer's server.

While the intervention participants will see the above described download instructions prior to this step, control group participants will be directed to the gift code page immediately after completing their baseline survey. At this gift code page all participants will be presented with instructions on how to get their electronic gift code (such as from Amazon) as a thank-you for their time. The amounts are \$25 for the baseline survey, \$25 for the 1-month survey, and \$50 for the 3-month survey. The Qualtrics software uses a Completely Automated Public Turing test to tell Computers and Humans Apart (CAPTCHA) to deter bots from claiming multiple gift cards.

The baseline survey and the 2 follow-up surveys will take about 40 minutes each to complete. The subject will be notified via email about when to complete the baseline, 1-month, and 3-month surveys. There will be an initial request to complete each survey, followed by 2 reminders (Appendix F).

#### Intervention.

Use. The consent form explains that the participant should spend about 30 minutes per week using the app, and that the average total estimated time to use the intervention over the 3-month study period is 6 hours. Regarding encouragement to use the app, within the app itself, there will be pop-up reminders about once per week to use various sections of the app during the 3-month study period.

Application content. Brief interventions (BI) are research-proven procedures for at-risk individuals to change substance abuse behaviors (USDHHS, 1999). Key elements of BI include screening or assessment, individualized feedback, addressing motivational underpinnings of the substance abuse, and teaching strategies for behavior change (Miller & Sanchez, 1994; USDHHS, 1999). Strong research evidence supports the effectiveness of brief interventions for substance users, particularly users identified in medical settings (Heather, 1995; Kahan et al., 1995; Mattick and Jarvis, 1994; Wilk et al., 1997). Although brief interventions are traditionally delivered face-to-face, evidence suggests that electronic delivery of these interventions may be an effective and efficient alternative. Self-assessment and provision of feedback are components of BI that are particularly amenable to electronic delivery.

As a patient-centered prevention effort, the Mobile Application for Prescription Drug-Abuse Education (MAPDE) is a brief intervention in a mobile phone app that focuses on enhancing critical communication and decision-making skills to help military members reduce prescription drug misuse. It contains modules to: (1) assess risk for medication misuse and related behavioral health concerns; (2) provide individualized feedback on risk level with recommendations to view related sections within the app; (3) store information on current medications and look up drug interaction and related information; (4) enhance critical communication and decision-making skills within healthcare and other interpersonal contexts by providing interactive virtual scenarios; (5) teach about the risks of prescription drug misuse; and (6) provide available resources for help with prescription drug misuse, all within an accessible mobile technology format. Screen shots of the final app will be provided to the IRB.

The app does not collect PHI or PII nor does it automatically transmit any PHI or PII to an external server, neither within the risk assessment module or elsewhere within the app. All

4

participant-entered responses to the questions in the app are contained within the smartphone itself. The app does contain an option for the user to send an email with information they've entered to their provider. This feature is to enhance communication between patient and provider regarding medication-relevant issues such as changes in medication side effects; however, it is completely the user's decision if and when to utilize the email feature, and what information to send.

Measures. The data collected for this study will be self-reported survey data collected at baseline, 1 month and 3 months after baseline (see surveys in Appendix G).

Risk of prescription drug misuse. Risk for prescription drug misuse will be measured using a 6-item scale previously used by Morasco and Dobscha (2008), which is actually a subset of the Pain Medication Questionnaire (PMQ) scale (Adams et al., 2004). The original scale was created to screen for prescription drug misuse among chronic pain patients undergoing opioid therapy, and the shortened scale was created for use among a military veteran population. The scale includes items such as: (1) At times I need to borrow pain medication from friends or family to get relief; and (2) How many times in the past year have you asked your doctor to increase your prescribed dosage of pain medication in order to get relief?

Additionally, the Current Opioid Misuse Measure (COMM) (Butler et al., 2007) will be used to measure risk for opioid prescription drug misuse. It measures 17 misuse behaviors over the past 30 days for those currently taking medications.

<u>Preparedness to talk about prescription drug misuse</u>. Four items assess the level of preparedness to talk to others about a personal concern for prescription drug misuse or a concern about others' possible misuse.

<u>Knowledge</u>. Twenty-three multiple choice knowledge items will assess the participant's level of knowledge of the definition of misuse and related educational points.

Attitudes. Forty-one attitudinal items will assess prescription drug misuse-related attitudes. Eight items came from the Prescription Drug Attitudes Questionnaire (PDAQ) (Bodenlos et al., 2014) and were adapted by the investigators for the military. Five items measure perceived harm (O'Neill, 2011), which were adapted from the Monitoring the Future study. There are 26 additional investigator-developed items that specifically align with the app's main messages. And finally, there are two additional items on perceived behavioral control indicating decisions to stay away from misusing and from abusing prescription drugs (O'Neill, 2011).

<u>Medication use and pain</u>. Seven yes/no items will assess current medication use, prescription medication use and pain medication use, as well as pharmacy use, injury or illness and current pain. Also, one item will assess the medication use of others in the participant's household.

Mental well-being. Because poorer psychological health is associated with higher risk for prescription medication misuse, 13 items will assess mental well-being. PTSD symptoms will be assessed using the Primary Care-PTSD scale (PC-PTSD) (Prins et al., 2003), which is a four-item subscale of the PTSD Checklist (Weathers, Litz, Herman, Huska, & Keane, 1993) with yes/no response options. Depressive and anxiety disorders will be measured with the brief Patient Health Questionnaire 4 (PHQ-4) for use in a general population (Kroenke, Spitzer, Williams, & Lowe, 2009). Two items are designed to detect the presence of depression and the other two items screen for generalized anxiety disorder. Traumatic brain injury (TBI) will be assessed with 3 items based on the Defense and Veterans Brain Injury Center TBI screening tool (Schwab, Baker, Ivins, et al., 2006).

Demographics. The baseline survey will have 10 items inquiring about the participant's

demographics such as age, sex, education, rank, race/ethnicity and branch of service, and military background questions on ever having been deployed and the total number of combat deployments. The demographic items closely match those in the National Center for Health Statistics annual survey.

<u>Usage and user ratings</u>. Experimental group participants only will receive 21 items about their experience with the app in the 1-month and 3-month surveys. These items will assess time spent using the app, ease of use, overall satisfaction with the app, usefulness of particular sections, relevance of the content, etc.

In addition, aggregated data on app page views and navigation information will be collected from the app developer's server. The information is collected securely and anonymously for post-study research analysis purposes. The app will be developed such that every entry and exit from any mobile app page creates a time-stamped event, which is transmitted to the app developer's server. The event information collected contains information on the page title, a time stamp, and event type (e.g., entry or exit). Using this collected data, analyses can be performed about the page view duration and navigation patterns. This data can also provide information on the number of times a page is visited during the study. The aggregated collected data can be viewed by the NHRC research staff during the study by logging into the developer's web portal. This aggregated data cannot be tracked back to individual users.

Statistical analysis plan. Results will be analyzed using a 2 x 3 (group: experimental/control, by time: baseline/1-month/3-month), repeated measures analyses of variance (ANOVA) to examine the potential effectiveness of the program over the 3-month study period. Categorical outcomes will be analyzed using generalized linear mixed models for binary outcomes. Group by time interactions will be examined for any evidence of improvement where greater positive changes in risk for misuse and related outcomes for the experimental group compared to the control group are observed. In addition, descriptive statistics will be used to assess the sample and to examine experimental group participants' satisfaction with and use of the app. Attrition analyses using independent t-tests and Chi-square tests will be carried out among the total sample, as well as by group to examine differences in participant characteristics among attriters and non-attriters. An alpha level of 5% will be assumed in all statistical tests. All analyses will be conducted using IBM SPSS Statistics 19.0.

#### 2. Sample Size Determination With Statistical Power Calculation

This study will determine if there is evidence that participants using the app will show greater positive change in their risk of prescription drug misuse and related outcomes compared to the control group over time. We calculated a minimum sample size based on analyzing the group by time interaction (2 groups (experimental, control) by 3 time points (baseline, 1 month, 3 month)) for a repeated measures ANOVA, using the software program G\*Power (Faul et al. 2007). The researchers are not aware of any previous evaluation of a prescription drug misuse prevention app. However, in a systematic review of electronicbased interventions that utilize behavior change techniques, the reported average effect size for health behavior change was small (about d=.20) (Webb et al., 2010). However, none of the interventions focused on the population of patients using pain medications and prescription drugs with risk for abuse. Considering that this population may be slightly more motivated, we used an effect size of f=.175, which is roughly equivalent to d=.35, which is still considered a small effect size. Given a small effect size (f) of .175 with a power level of .80, a desired significance level of .05, an estimated correlation between time points of .5, and assuming a two-tailed test, our required total sample size is 54. Thus, we have set our goal for 60 participants to complete the full study as this should be adequate to provide the statistical power to examine evidence of differential effects between groups and to estimate effect sizes. Given an estimated 25% attrition rate over the 3-month study period, we plan to initially enroll 80 participants, which would then be reduced to a final sample of 60 participants for analysis.

#### 3. Justification for Exclusion of Specific Groups

Non-active duty personnel, service members younger than age 18, personnel in a service branch other than the Navy or Marine Corps, persons reporting that they do not have a smartphone, and those not currently taking a prescription medication with the potential for abuse will be excluded. The first three are excluded for regulatory purposes and the final two because of the nature of the product being evaluated.

#### 4. Required Equipment and Supplies

Researchers will use computers, smartphones, telephones and general office supplies for conduct of the work related to this protocol.

#### VII. ORGANIZATION OF RESEARCH EFFORT

#### 1. Duties and Responsibilities

Suzanne Hurtado will serve as the Principal Investigator. She will be responsible for the overall conduct of the study including day-to-day operation of the study, subject recruitment, consenting procedures, collecting data, data analyses, and writing.

Co-investigator, Cynthia Simon-Arndt, will be responsible for assisting with subject recruitment and consenting procedures, collecting data, addressing and coordinating technical issues related to the app, and co-writing the report.

Co-investigator, Cynthia Thomsen, will conduct the statistical analyses and assist with co-writing the report.

Associate investigator, Stephanie Kewley, will conduct the statistical analyses and assist with co-writing the report.

Key support - Ms. Renee Dell'Acqua will be responsible for assisting with the day-to-day operation of the study and data management.

Key support - Ms. Elizabeth Lauer, Ms. Robyn Martin, Ms. Shannon Fitzmaurice and Mr. Casey Kohen will be responsible for assisting with subject recruitment and preparing emails for recruited subjects.

The technology developers (Intelligent Automation, Inc.) will provide the revised version of the app for the test. They will not interact with any subjects and they will not have access to any identifiable data. They will receive the final report from this study.

All investigators involved with subjects or their data in this study have completed HIPAA and NHRC IRB/Ethics training.

#### 2. Chain of Command

All of the co-investigators and key support personnel (Cynthia Simon-Arndt, Cynthia Thomsen, Renee Dell'Acqua, Robyn Martin, Elizabeth Lauer, Casey Kohen, and Shannon Fitzmaurice) will report directly to the Principal Investigator, Suzanne Hurtado.

#### VIII. RISKS AND DISCOMFORTS TO RESEARCH VOLUNTEERS

#### I. Risk to the Volunteer and Means of Mitigation

The main potential risk is the small chance of accidental disclosure, or breach of confidentiality, of the participants' survey responses. The primary means of mitigation of accidental disclosure of a participant's

7

security, passwords, and encryption, in compliance with DoDD 8500.01E and DoDI 8500.2 instructions; (3) transferring all survey data from Qualtrics to a secure server at Naval Health Research Center and deleting all survey data from the Qualtrics server once a month throughout the study data collection period; (4) not storing respondents' IP addresses as the survey data are received; (5) not storing respondents' phone ID number with the summary usage data; (6) using the app developer's secured SSH and SSL 128-bit encrypted server to collect the aggregated, summary usage data, and for the PI to enter the web portal to create a unique key number for participants; (7) storing all electronic data using password protected files on a secure server at Naval Health Research Center (NHRC); (8) keeping all paper copies of any data in locked files at NHRC; (9) immediately deleting email addresses from the data after all surveys have been linked; and (10) limiting access to all data to approved-investigators involved in this study.

Regarding information that participants enter into the smartphone app, none of this information will contain personal identifiers. Furthermore, this information will not automatically be sent to any server; it will only be housed on the participant's personal smartphone. Instructions provided to the user will encourage them to protect access to their phone by setting up a PIN. In addition, participants will be advised that they further protect their phone by not allowing automatic Wi-Fi connections to unknown devices or networks. The app contains a feature where the user can opt to email information from the app on their phone to their physician, but this feature will be clearly designated as optional; the participant decides if they want to share any information and what that information is.

Another possible risk is that participants may find it uncomfortable to address prescription drug misuse and related psychological and behavioral health issues. The primary means of mitigating this risk is that within the app, they do not have to answer any questions that they do not want to. Also, while the researchers recommend that the participant use the app for a certain number of hours, the participant is in control of how much or how little they use the app. Regarding the surveys, participants will be informed that they don't have to answer any questions that they don't want to and that they may stop at any time. In addition, participants will be provided with the phone number to the Veteran's Crisis Center in the consent form and within the app, which they may choose to contact for assistance in the event that their participation causes them discomfort and/or they feel an urgent need for behavioral health assistance.

#### 2. Special Risks to Pregnant Women

There are no known special risks to pregnant women related to this study.

#### 3. Safety Precautions and Emergency Procedures

Aside from in-person recruitment efforts, this study involves phone and email contact and is primarily a web-based study. In the unlikely event that an unexpected emergency arises during in-person interaction with the potential subject, it would be onsite at the hospital and the study staff will alert appropriate hospital staff for immediate medical attention for the research participant, if necessary. If an emergency arises at any other time during the conduct of this study, participants will have been advised in the consent form that they should call 911 or their local emergency medical services for help.]

#### 4. Assessment of Sufficiency of Plans to Deal With Untoward Events or Injuries

The use of standard Navy medical procedures has been deemed sufficient to deal with any untoward events and/or injuries. These procedures include alerting appropriate hospital staff for immediate medical attention for the research participant, if necessary, when the study staff is interacting with the participant in person at NMCSD. In all other situations, the participant shall call 911 or their local emergency medical services for help.

#### 5. Qualification Research Monitor and Medical Support Personnel

N/A

#### IX. DESCRIPTION OF THE SYSTEM FOR MAINTENANCE OF RECORD

#### 1. Experimental Data

This study will collect private health information and personal email address (an element that the Department of Navy, Chief Information Officer, considers as personally identifiable information (PII), DON CIO, 2011; and is Protected Health Information (PHI)). Subject privacy and data confidentiality will be maintained through the procedures described above in the Risk section and below.

Paper records will be kept in locked filing cabinets at Naval Health Research Center (NHRC), Barracks Building 328, Rm. 205A, with access limited to the IRB-approved investigators involved in this study. All electronic data will be stored using password protected files on a secure server at NHRC. Access to all electronic data will be limited to the IRB-approved investigators involved in this study. The information obtained will be used only by study personnel. The paper records and electronic information obtained in this study will be maintained for three years after the primary study results have been provided to the funding sponsor. Participant emails will be deleted from files after surveys have been matched and the data collection is complete. Data will be used for immediate analyses conducted by the researchers at NHRC. No personally identifiable information will be used by or disclosed (released) to another institution.

The summary results of this study will be presented to the military medical treatment facility that provides access to the potential participants, the technology development partners at Intelligent Automation, Inc., and to the sponsor, the National Institute on Drug Abuse (NIDA). The summary results may also be published in Department of Defense technical reports, scientific journals, or presented at scientific meetings. No publication or presentation about the research study will reveal a participant's identity. Only overall statistics such as averages and percentages for the group will be presented; no study results will be reported for individuals. Lastly, individuals from official government agencies, such as the Department of Defense, US Navy, and US Army, may inspect the research records to ensure that the rights and safety of all research participants are protected.

2. Research Protocol, Consent Forms, and Related Documents for Protection of Human Research Volunteers

The principal investigator will keep the research protocols and consent forms in a locked file in Bldg. 328, Room 205A.

3. Individual Medical Records

No official medical records will be accessed for this study.

4. Conflict of Interest

No person involved in the design, conduct, or reporting of this research has a financial or other interest that could reasonably appear to be affected by the carrying out or the results of this research.

X. APPENDICES

Evaluation of a Mobile Application for Prescription Drug Abuse Education

#### A. VOLUNTARY CONSENT TO PARTICIPATE IN A RESEARCH STUDY

You are being asked to volunteer to participate in a research study called "Evaluation of a Mobile Application for Prescription Drug Abuse Education" (Protocol # NHRC.2016.0019). Taking part in this study is your choice. If you don't understand any part of this Consent Document, ask the investigators to explain that part of the study. If you have any questions, please ask any of the study staff.

Why is this study being done? The study will test a new smartphone application (an "app") to educate about prescription drug misuse. The app was made to help military members reduce their risk of prescription drug misuse. Researchers from Naval Health Research Center in San Diego, California will conduct the study. About 60 to 80 people recruited from a military medical treatment facility will take part in this research. We are asking you to take part in this study because you currently have a prescription for a medication with the potential for misuse. To take part in the study, you must be: (1) age 18 or over; (2) on active duty; (3) have a current prescription for a medication with the potential for misuse; and (4) own a smartphone.

What will happen if you decide to take part in this study? You will be asked to complete an online survey about prescription drug use, knowledge and attitudes related to prescription drug misuse, and mental well-being. The survey will happen at 3 points in time (an initial survey; 1 month later; and 3 months later). Your participation <u>must</u> be during your off-duty time. Each survey will take about 40 minutes to complete. We will ask for your personal email address to contact you about the study and to link your surveys over time.

You will be randomly assigned to: (1) use the smartphone app for this study and continue with your physician's care and treatment as usual; or (2) continue with your physician's care and treatment as usual (no smartphone app). The app contains various educational sections and tools such as: self-assessments for risk of misuse with tailored feedback and recommendations; information on misuse, drug interactions and more; scenarios to practice communication skills related to preventing misuse; resources for help and more. If you are assigned to use the app, we request that you use the app for at least 30 minutes per week for a 3-month period (which would be a total of about 6 hours over a 3-month study period). If you are not assigned to use the app, you will still receive a list of resources for help with prescription drug and other substance abuse issues. Whichever group you are in, this study will not interfere in any way with your usual medical treatment.

We will not use your name in the study, but we will ask for your non-DoD (personal) email address to communicate with you about the study and you will enter your email address in the online surveys. At the end of the study we will delete your email address from our files. We encourage you to create a new email address that does not contain any identifying information for this study.

What are the risks if you take part in this study? The investigators believe that the risks or discomforts to you from participating in this study are minimal. One possible risk is that you may find it uncomfortable to answer survey questions or app assessment questions, or that the topic of prescription drug misuse and related psychological and behavioral health issues may make you uncomfortable. You don't have to answer any questions in the surveys or in the app that you don't want to, and you can stop participating at any time. If you feel that you are experiencing distress from this study, please call the Veterans Crisis Line (800-273-8255). If you need emergency medical help at any time during the conduct of this study, call 911 or your local emergency medical services for help.

Another possible risk is the slight risk of accidental disclosure of your survey answers and personal email address. The study staff will protect the data that is collected in this study. Your email will not be used for any other purpose. Furthermore, emails will be deleted from the researchers' files immediately after the data collection is complete. Safeguards listed below are in place to protect the confidentiality of your information.

Another possible risk is that someone may look at your responses to the app on your smartphone. For this reason we encourage you to use safe handling practices for your phone such as not leaving it unattended and using a PIN to lock it. Responses you enter into the app are not automatically sent to any server; they will only be housed on your smartphone. It is your decision if you would like to email any information from the app to someone else—your doctor, for example. In addition, we will be collecting usage data from the app developer's secure server, but this usage data will be anonymous; it will not be linked with your phone ID number or any other personally identifying information.

What happens if you have a medical problem while you take part in this study? If you are injured or become ill because of taking part in this study, call 911 or your local emergency medical services for emergencies, or contact your doctor for help. Also, please contact the study Principal Investigator, Suzanne Hurtado, at (619) 607-1910 or <a href="mailto:suzanne.l.hurtado.civ@mail.mil">suzanne.l.hurtado.civ@mail.mil</a>, or the IRB Chairman, William Becker, at (619) 553-8424 or <a href="mailto:USN.NHRC.IRB@mail.mil">USN.NHRC.IRB@mail.mil</a> to inform them of the problem. By indicating your consent on this form, you will not be giving up any legal rights.

Are there benefits to taking part in this study? You won't receive any direct benefit from taking part in this study, but the information gained from this study may help researchers learn more about how to best prevent prescription drug misuse. This could ultimately help service members in the future.

Will you be compensated for participating in this study? As a thank-you for your participation, you will be emailed Amazon gift codes in the amount of \$25 for the initial survey; \$25 for the 1 month survey; and \$50 for the 3 month survey. Your participation must be during off-duty, liberty or leave status in order to be compensated for participating in the study.

What health information will be collected and will it be kept confidential to the extent permitted by law? If you choose to take part in this study, the online surveys and the self-assessments within the app will ask you questions about prescription drug use, knowledge and attitudes related to prescription drug misuse, and mental well-being. All survey data you provide online will be collected with your personal email address; we will delete your email address from our files at the end of the study. No other data that you enter into the app itself is being collected. You will not be asked to disclose identifiable personal medical information.

In addition, we will be collecting usage data from the app developer's secure server. This usage data will be anonymous; it will not be linked with your phone ID number or any other personally identifying information.

The information from the study will be used only by study staff and will be held in confidence. No one in your chain-of-command or at your command will ever see your survey answers. Surveys will be completed over the Internet on a server that uses a high-end firewall system, transport layer security, passwords, and encryption.

To further help protect your privacy, we have obtained a **Certificate of Confidentiality** from the National Institutes of Health. The researchers can use this Certificate to legally refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below. As described above, the only personally identifying information we are using is your personal email address.

The Certificate cannot be used to resist a demand for information from personnel of the United States Government that is used for auditing or evaluation of federally funded projects. You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers may not use the Certificate to withhold that information.

In addition, while your survey responses will be protected as described above, your verbal comments to the researchers are not. Therefore, if you voluntarily tell the researchers of any intention to do harm to another person, or to yourself, or indicate child abuse, the researchers may have to report this to the appropriate authorities (suicide crisis center or military police, for example). The Certificate of Confidentiality will not be used to prevent such disclosures.

Ms. Suzanne Hurtado is responsible for storing the information collected from the study. This information will be protected by keeping all paper records in locked files in building 328 at Naval Health Research Center. Electronic data will be stored using a password protected files on a secure server at Naval Health Research Center. Access to all data will be limited to staff involved in this study. No personally identifying information will be used by or disclosed (released) to another institution.

You may change your mind and revoke (take back) your permission to collect or use your information at any time. To revoke your permission, please write to Ms. Suzanne Hurtado at suzanne.l.hurtado.civ@mail.mil. When you revoke your permission, no new health information about you will be gathered after that date and you may no longer be allowed to participate in the study. Information that has already been gathered will be removed from the electronic database for this study, if your personal email address has not already been deleted.

The summary results of this study will be presented to the medical treatment facility involved in the research, the technology development company (Intelligent Automation, Inc.), and to the National Institute on Drug Abuse. The results may also be published in Department of Defense technical reports, scientific journals, or presented at scientific meetings. No publication or presentation about the research study described above will reveal your identity. Only overall statistics such as averages and percentages for groups will be presented; no study results will be reported for individuals. Lastly, individuals from official government agencies, such as the Department of Defense, US Navy, and US Army, may inspect your research records to ensure that the rights and safety of all research participants are protected.

What are your rights if you take part in this study? Taking part in this study is your choice. Your participation must be completely voluntary. If you decide to take part, you may still leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any benefit to which you are otherwise entitled.

What if you have questions about the study? Make sure that you have had a chance to ask questions and have received satisfactory answers to all of your questions. You should contact the following individuals to answer your questions:

For questions about the research, contact Suzanne Hurtado at (619) 607-1910 or suzanne.l.hurtado.civ@mail.mil.

For questions about the ethical aspects of this study or subjects' rights, contact William Becker at (619) 553-8424 or USN.NHRC.IRB@mail.mil. He is the Chairman of the Naval Health Research Center Institutional Review Board, a group of people who review the research to protect your rights.

#### CONSENT TO TAKE PART IN THIS RESEARCH STUDY

By clicking on the "I consent" box below, you indicate that you have read the information in this form and have had a chance to ask any questions you have about the study and its procedures and risks, as well as any of the other information contained in this consent form. All of your questions have been answered to your satisfaction. You understand that this is research. Your clicking on the "I consent" box also indicates that you voluntarily agree to be in this research study and understand that you can change your mind and withdraw your consent to participate at any time. You authorize the use of the survey data and app usage data as described in this consent document.

| Ple | ase check one: |
|---|---|
| | I consent to participate in this research study. |
| | I DO NOT consent to participate in this research study. |
| Plea | ase indicate agreement with the statement below by checking the box. |
| | I attest that I am participating in this study while in off-duty, liberty or leave status. |

#### **PRIVACY ACT STATEMENT**

**AUTHORITY:** 

32 CFR Part 219, Protection of Human Subjects; 45 CFR Part 46, Protection of Human Subjects; DoDI 3216.02, "Protection of Human Subjects and Adherence to Ethical Standards in DoD-Supported Research," October 20, 2011; 45 CFR Parts 160 and 164, Health Insurance Portability and Accountability Act (HIPAA) Privacy and Security Rules; and E.O. 9397 (SSN), as amended. License to administer this survey is granted per OPNAVIST 5300.8C under OPNAV Report Control Symbol 6320-5, which expires 28FEB2020, and under Marine Corps SCN USMC-IR-17002.

**PURPOSE:** 

Information is collected to enhance basic medical knowledge, or develop tests, procedures, and equipment to improve diagnosis, treatment, or prevention of illness, injury, or performance impairment under research protocol NHRC.2016.0019, titled "Evaluation of a Mobile Application for Prescription Drug Abuse Education."

**ROUTINE USES:** 

In addition to those disclosures generally permitted under 5 U.S.C. 552a(b) of the Privacy Act of 1974, the DoD "Blanket Routine uses" under 5 U.S.C. 552a(b)(3) apply to this collection. Medical research information will be used for analysis and reports by the Department of the Navy and Defense, and other U.S. Government agencies, provided this use is compatible with the purpose for which the information was collected. Use of the information may be granted to non-Government agencies or individuals by the Navy Surgeon General following the provisions of the Freedom of Information Act or as may be indicated in the accompanying Informed Consent Form.

DISCLOSURE:

Provision of information is voluntary. There are no penalties for not providing requested information, but failure to provide the requested information may result in failure to be accepted as a research volunteer in an experiment or removal from the program.

#### **B. INVESTIGATOR COMPLIANCE ATTESTATION**

Cianaturas and datas:

#### INVESTIGATOR COMPLIANCE ATTESTATION

As a researcher or team member responsible for performing and monitoring the research under the protocol titled Evaluation of a Mobile Application for Prescription Drug Abuse Education, I have read and understand the provisions of Title 32 Code of Federal Regulations Part 219 (Protection of Human Subjects), Department of Defense (DoD) Instruction 3216.02 (Protection of Human Subjects in DoD-Supported Research), DoD Instruction 6025.18-R (Privacy Rule), SECNAV Instruction 3900.39D (Human Research Protection Program), OPNAV Instruction 5300.8C (Personnel Surveys), NAVHLTHRSCHCEN Instruction 3900.2G (Protection of Human Subjects), NAVHLTHRSCHCEN Notice 6500 (Protection of Health Information in Research), Title 21 Code of Federal Regulations Parts 50, 56 if applicable (clinical investigations regulated by the FDA), and all relevant local instructions. I have disclosed all potential and actual conflict of interest(s) related to the design, conduct, analysis, or reporting of this research. I will abide by all applicable laws and regulations, and I agree that in all cases, the most restrictive regulation related to a given aspect of research involving protection of research volunteers will be followed. In the event that I have a question regarding my obligations during the conduct of this Navy-sponsored project, I have ready access to each of these regulations, as either my personal copy or available on file from the Chairperson of the Institutional Review Board. I understand that my immediate resource for clarification of any issues related to the protection of research volunteers is the Chairperson of the Institutional Review Board.

| Signatures and dates. | (DD/MM/11) |
|---|---|
| Correct Months MDH | // |
| Suzanne L. Hurtado, MPH Principal Investigator, Naval Health Research Center | |
| Cynthia M. Simon-Arndt | / |
| Co-Investigator, Leidos Inc., Naval Health Research Center | , |
| Cynthia Thomsen | |
| Co-Investigator, Naval Health Research Center | |
| Renee Deil'Acqua | // |
| Key Support, Leidos Inc., Naval Health Research Center | |

Version Date: 14 MAY 2018 B-1

#### INVESTIGATOR COMPLIANCE ATTESTATION

#### INVESTIGATOR COMPLIANCE ATTESTATION

As a researcher or team member responsible for performing and monitoring the research under the protocol titled Evaluation of a Mobile Application for Prescription Drug Abuse Education, I have read and understand the provisions of Title 32 Code of Federal Regulations Part 219 (Protection of Human Subjects), Department of Defense (DoD) Instruction 3216.02 (Protection of Human Subjects in DoD-Supported Research), DoD Instruction 6025.18-R (Privacy Rule), SECNAV Instruction 3900.39D (Human Research Protection Program), OPNAV Instruction 5300.8C (Personnel Surveys), NAVHLTHRSCHCEN Instruction 3900.2G (Protection of Human Subjects), NAVHLTHRSCHCEN Notice 6500 (Protection of Health Information in Research), Title 21 Code of Federal Regulations Parts 50, 56 if applicable (clinical investigations regulated by the FDA), and all relevant local instructions. I have disclosed all potential and actual conflict of interest(s) related to the design, conduct, analysis, or reporting of this research. I will abide by all applicable laws and regulations, and I agree that in all cases, the most restrictive regulation related to a given aspect of research involving protection of research volunteers will be followed. In the event that I have a question regarding my obligations during the conduct of this Navy-sponsored project, I have ready access to each of these regulations, as either my personal copy or available on file from the Chairperson of the Institutional Review Board. I understand that my immediate resource for clarification of any issues related to the protection of research volunteers is the Chairperson of the Institutional Review Board.

| | (DD/MM/YY) |
|------|------------|
| -,- | // |
| | // |
| 7.16 | // |

Version Date: 14 MAY 2018 B-2

#### C. REFERENCES

- Adams, L. L., Gatchel, R. J., Robinson, R. C., Polatin, P., Gajraj, N., Deschner, M., & Noe, C. (2004). Development of a self-report screening instrument for assessing potential opioid medication misuse in chronic pain patients. *Journal of Pain and Symptom Management*, 27(5), 440-459.
- American Forces Press Service. DOD Awards Contract for Device Management System, App Store. [Internet]. 2013; <a href="http://www.defense.gov/news/newsarticle.aspx?id=120388">http://www.defense.gov/news/newsarticle.aspx?id=120388</a>. Accessed February 13, 2014.
- Bodenlos, J. S., Malordy, A., Noonan, M., Mayrsohn, A., & Mistler, B. (2014). Prescription Drug Attitudes Questionnaire: Development and Validation. *Psychology*, 5(14), 1687-1693.
- Bray RM, Pemberton MR, Hourani LL, et al. 2008 Department of Defense Survey of Health Related Behaviors Among Active Duty Military Personnel: A component of the Defense Lifestyle Assessment Program (DLAP). Research Triangle Park, NC: Research Triangle Institute; 2009. 10940-FR.
- Bray RM, Pemberton MR, Lane ME, Hourani LL, Mattiko MJ, Babeu LA. Substance use and mental health trends among U.S. military active duty personnel: Key findings from the 2008 DoD Health Behavior Survey. *Military Medicine*. 2010;175(6):390-399.
- Butler SF, Budman SH, Fernandez KC, Houle B, Benoit C, Katz N, Jamison RN. Development and validation of the Current Opioid Misuse Measure. *Pain.* 2007;130:144-156.
- Department of the Navy (2015). Health of the Force Report.
- Faul F, Erdfelder E, Lang A-G, Buchner A. (2007). G\*Power 3: A flexible statistical power analysis program for the social, behavioral, and biomedical sciences. *Behavior Research Methods*, 39, 175-191.
- Friedman RA. Wars on Drugs. [Internet]. 2013; http://www.cchrint.org/2013/04/08/ny-times-wars-on-drugs/. Accessed April 13, 2013.
- Heather N. Interpreting the evidence on brief interventions for excessive drinkers: The need for caution. *Alcohol and Alcoholism*. 1995;30(3):287–296.
- Kahan M, Wilson L, Becker L. Effectiveness of physician-based interventions with problem drinkers: A review. Canadian Medical Association Journal. 1995;152(6):851-859.
- Kroenke K, Spitzer R, Williams JW, Lowe B: An ultra-brief screening scale for anxiety and depression: the PHQ-4. *Psychosomatics*. 2009;50(6): 613–21.
- Mattick RP, Jarvis T. Brief or minimal intervention for 'alcoholics'? The evidence suggests otherwise. Drug and Alcohol Review. 1994;13:137-144.
- Miller WR, Sanchez VC. Motivating young adults for treatment and lifestyle change. Howard GS. (Ed), Nathan PE (Ed), (1994). Alcohol use and misuse by young adults. (pp. 55-81). Notre Dame, IN, US: University of Notre Dame Press, vi, 198 pp.
- Morasco BJ, Dobscha SK. Prescription medication misuse and substance use disorder in VA primary care patients with chronic pain. *General Hospital Psychiatry*. 2008;30(2):93-99.
- O'Brien CP, Oster M, Morden E. Substance Use Disorders in the U.S. Armed Forces. Washington, DC: Committee on Prevention, Diagnosis, Treatment and Management of Substance Use Disorders in the U.S. Armed Forces, National Academy of Sciences, Institute of Medicine; 2012.
- O'Neill, AK. "Norms, Attitudes, Perceptions, and Intentions for Benzodiazepine Prescription Drug Abuse Among Adolescents" (2011). Master's Theses and Doctoral Dissertations. Paper 422.
- Prins A, Ouimette P, Kimerling R, Cameron RP, Hugelshofer DS, Shaw-Hegwer J, ... Sheikh JI. (2003). The primary care PTSD screen (PC-PTSD): development and operating characteristics. *Primary Care Psychiatry*, 9(1), 9-14.

Version Date: 14 MAY 2018 C-1

- Schwab K, Baker G, Ivins B, Sluss-Tiller M, Lux W, Warden D. (2006). The Brief Traumatic Brain Injury Screen (BTBIS): Investigating the validity of a self report instrument for detecting traumatic brain injury (TBI) in troops returning from deployment in Afghanistan and Iraq. *Neurology*, 66, A235.
- U.S. Department of Health and Human Services. Brief Interventions and Brief Therapies for Substance Abuse, *Treatment Improvement Protocol (TIP) Series, No. 349*. Center for Substance Abuse Treatment report, DHHS Report No. (SMA) 99-3353. Rockville, MD: Substance Abuse and Mental Health Services Administration; 1999.
- Weathers FW, Litz BT, Herman DS, Huska JA, Keane TM. (1993, October). The PTSD Checklist (PCL): Reliability, validity, and diagnostic utility. Paper presented at the annual meeting of the International Society of Traumatic Stress Studies, San Antonio, TX. Retrieved from <a href="http://www.pdhealth.mil/library/downloads/pcl sychometrics.doc">http://www.pdhealth.mil/library/downloads/pcl sychometrics.doc</a>.
- Webb TL, Joseph J, Yardley L, Michie S. Using the internet to promote health behavior change: a systematic review and meta-analysis of the impact of theoretical basis, use of behavior change techniques, and mode of delivery on efficacy. *Journal of Medical Internet Research*, 2010;12(1), doi: 10.2196/jmir.1376.
- Webster LR, Webster RM. Predicting aberrant behaviors in opioid-treated patients: preliminary validation of the opioid risk tool. *Pain Medicine*, 2005;6(6):432-442.
- Wilk AI, Jensen NM, Havighurst TC. Meta-analysis of randomized control trials addressing brief interventions in heavy alcohol drinkers. *Journal of General Internal Medicine*. 1997;12(5):274–283.
- Zoroya G. Abuse of pain pills by troops concerns Pentagon. [Internet]. 2010; http://usatoday30.usatoday.com/news/military/2010-03-16-military-drugs\_N.htm. Accessed April 13, 2012.

Version Date: 14 MAY 2018 C-2

#### D. LIST OF MEDICATIONS

#### Prescription Drugs with the Potential for Misuse

Abstral oxycodone, acetaminophen oxycodone hydrocholide. acetaminophen codeine phosphate, acetaminophen hydrocodone bitartrate, acetaminophen Actiq alprazolam Ambien CR Amrix Ascomp with Codeine carisoprodol, aspirin, codeine phosphate oxycodone, aspirin Ativan diphenoxylate hydrochloride, atropine sulfate Belsomra Bupap butabarbital sodium Butalbital Carbatrol carisoprodol carisoprodol, aspirin Cheratussin AC chloral hydrate codeine phosphate, chlorcyclizine chlordiazepoxide chlorzoxazone clonazepam clorazepate codeine phosphate codeine phosphate. guaifenesin codeine phosphate, promethazine Codeine Sulfate cyclobenzaprine Dalmane Diastat diazepam Dolophine Donnatal Lorcet Plus

doxepin hydrochloride Duragesic Edluar Endodan Esgic estazolam eszopiclone Exalgo fentanyl fentanyl buccal fentanyl citrate Fioricet Fioricet with Codeine **Fiorinal** Fiorinal with Codeine Fexmid flurazepam flurazepam hydrochloride Halcion hydrocodone bitartrate, homatropine methylbromide hydrocodone Polistirex, chlorpheniramine Polistirex hydrocodone bitartrate, chlorpheniramine maleate, pseudoephedrine hydrochloride hydrocodone hydromorphone hydromorphone hydrochloride Indocin indomethacin Intermezzo Klonapin Lazanda Librax Librium Lomotil lorazepam Lorcet Lorcet HD

Lunesta meperidine meperidine hydrochloride meprobamate metaxalone methadone hydrochloride methocarbamol midazolam Nembutal Niravam Norco Norflex Norgesic Norgesic Forte Onsolis Opana Opana ER orphenadrine citrate orphenadrine citrate, aspirin, caffeine oxazepam Oxecta Oxycet oxycodone oxycodone HCL oxycodone Hydrochloride oxycodone hydrochloride, acetaminophen Oxycontin oxymorphone oxymorphone hydrochloride Palladone Parafon Forte DSC pentobarbital Percocet Percodan Phenobarbital Phrenilin Placidyl Promethazine VC with Codeine ргорохурнене Prosom quazepam ramelteon Reprexain

Restoril

Doral

Lortab

## Hurtado, Evaluation of a Drug Abuse Educational App, Protocol # NHRC.2016.0019

Rezira Robaxin Roxicet Roxycodone Rozerem secobarbital Seconal Silenor Sinequan Skelaxin Soma

Somnote Sonata Sublimaze Subsys suvorexant Synalgos Targiniq ER temazepam Tivorbex Tranxene triazolam Tussicaps

Tussionex Pennkinetic Tylenol 3 Tylenol 4 Tylenol with Codeine

Valium

Vicodin Vicoprofen Vituz Xanax Xartemis XR zaleplon zebutal Zohydro zolpidem

zolpidem tartrate **Zolpimist** Zutripro

#### E. FLYER

# Attention service members currently taking a prescription medication

# Do you enjoy using smartphone apps?

Naval Health Research Center is conducting a study to test an educational app on preventing prescription medication misuse.

Qualified participants will receive gift cards as a thank-you.

We will request your non-DoD email address to participate in this study. All information will be kept private and confidential.

# Contact us today for more information!

(619) 607-1910 or email: <a href="mailto:suzanne.l.hurtado.civ/@mail.mil">suzanne Hurtado, Principal Investigator</a>
Evaluation of a Mobile Application for Prescription Drug Abuse Education (NHRC IRB Protocol # NHRC.2016.0019)
Naval Health Research Center, San Diego, CA

 Evaluation of a Mobile Application for Prescription Drug Abuse Education (MNIRC.2015.0019) Call or text Suzanne Hurtado, Principal Investigator, 619 607-1910 or email: suzanne. Lhurtado.cdv@mail.mil Navol Health Research Center, San Diego, CA

Evaluation of a Mobile Application for Prescription Drug Abuse Education (#NHRC\_2016.0019)
Call or text Suzanne Hurlado, Principal Investigation et al. 9607-1910 or email: suzanne. Lhurtado, dw@mail.mil Navat Health Research Center, San Diego, CA

Evaluation of a Mobile Application for Prescription Drug Abuse Education (#NHRC\_2016.0019)
Call of text Suzanne Hutado, Principal investigator, 619 607-1910
or emali: suzanne. I.hurado. civ@mail..mil
Naval Health Research Center, San Diego, CA

Evaluation of a Mobile Application for Prescription
Drug Abuse Education (#NHRC.2016.0019)
Call or text Suzanne Hurtado, Principal Investigator
619-607-1910
or email: suzanne Lhurtado.ctw@mail.mil
Maxall Health Research Center San Dieso, CA

#### F. SURVEY INVITATIONS AND REMINDERS

#### **Baseline Survey Invitation Email**

Dear study participant,

Thank you for your interest in this study on the prevention of prescription medication misuse. Please see the attached consent form for the study.

Using a non-military mobile device or computer, please go to our study website: http://XXX to get started. If you decide to participate, please fill-out the first survey for this study and submit it within the next three (3) days. The information you provide will be kept completely confidential.

The study website asks you to enter your non-DoD (personal) email address. If you would like to create a new personal email address and account on Gmail for this study – one that does not contain any part of your name or other potentially identifying information – follow the instructions below.

- On your mobile device, open up your internet browser and go to the Google home page; https://www.google.com/
- 2. Click on Gmail at the top right corner of the page.
- 3. Click "Create an account".
- 4. Fill in the requested information. This includes 'choose your username'. This is the unique email address that you wish to use, which will be placed before '@gmail.com'. Because it needs to be unique, Google may have to check the availability of any name that you decide on to make sure that no one already has it.
- 5. Create a password.
- 6. 'Prove you're not a robot' by typing in the text that you see on the screen.
- 7. Click the box if you agree to the Google Terms of Service and Privacy Policy. Then click "Next step".
- 8. Click "Next step", then "Add Profile Photo" if you like, then "Next step" again to complete setting up your email.

Then send your new email address to the PI at Suzanne.l.hurtado.civ@mail.mil so we know how to contact you.

As a thank you, when you submit your survey, you will receive \$25.00 in e-gift codes within approximately 2 business days. As a reminder, you must participate during off-duty, liberty or leave status if you wish to be compensated.

If you have any questions about the study, or if you do not wish to participate or be contacted any more, please contact Suzanne Hurtado at Suzanne.l.hurtado.civ@mail.mil, or (619) 607-1910.

Thanks!
Suzanne Hurtado
Principal Investigator
Evaluation of a Mobile Application for Prescription Drug Abuse Education (#NHRC.2016.0019)
Naval Health Research Center, San Diego, CA
(619) 607-1910, Email: Suzanne.l.hurtado.civ@mail.mil

#### **Baseline Survey Reminder Email**

Dear study participant,

Thank you for your interest in this study on the prevention of prescription medication misuse. If you have already completed the first survey for this study, thank you and please disregard this email. If you have not completed the first survey, please see the attached consent form for the study.

Using a non-military computer, please go to our study website: http://XXX to get started. If you decide to participate, please fill-out the first survey for this study and submit it within the next three (3) days. The information

APPROVED

DATE: 6 14 1 18

EXP: 6 14 1 19

you provide will be kept completely confidential.

The study website asks you to enter your non-DoD (personal) email address. If you would like to create a new personal email address and account on Gmail for this study – one that does not contain any part of your name or other potentially identifying information – follow the instructions below.

- 1. On your mobile device, open up your internet browser and go to the Google home page: https://www.google.com/
- 2. Click on Gmail at the top right corner of the page.
- 3. Click "Create an account".
- 4. Fill in the requested information. This includes 'choose your username'. This is the unique email address that you wish to use, which will be placed before '@gmail.com'. Because it needs to be unique, Google may have to check the availability of any name that you decide on to make sure that no one already has it.
- 5. Create a password.
- 6. 'Prove you're not a robot' by typing in the text that you see on the screen.
- 7. Click the box if you agree to the Google Terms of Service and Privacy Policy. Then click "Next step".
- 8. Click "Next step", then "Add Profile Photo" if you like, then "Next step" again to complete setting up your email.

Then send your new email address to the PI at Suzanne.l.hurtado.civ@mail.mil so we know how to contact you.

As a thank you, when you submit your survey, you will receive \$25.00 in e-gift codes within approximately 2 business days. As a reminder, you must participate during off-duty, liberty or leave status if you wish to be compensated.

If you have any questions about the study, or if you do not wish to participate or be contacted any more, please contact Suzanne Hurtado at Suzanne.l.hurtado.civ@mail.mil, or (619) 607-1910.

Thanks!
Suzanne Hurtado
Principal Investigator
Evaluation of a Mobile Application for Prescription Drug Abuse Education (#NHRC.2016.0019)
Naval Health Research Center, San Diego, CA
(619) 607-1910, Email: Suzanne.l.hurtado.civ@mail.mil

DATE: 6 14 118
EXP: 6 114 119
Naval Health Research Center San Diego

#### 1-Month Survey Invitation Email

Dear study participant,

About one month ago you filled out a survey about the prevention of prescription medication misuse. Thanks for your participation! We now request that using a non-military mobile device or computer, you go to our study website: http://XXX and fill-out the 1-month survey for this study. Please submit it within the next three (3) days. The information you provide will be kept completely confidential.

As a thank you, when you submit this survey, you will receive \$25.00 in e-gift codes within approximately 2 business days. As a reminder, you must participate during off-duty, liberty or leave status if you wish to be compensated.

If you have any questions about the study, or if you do not wish to participate or be contacted any more, please contact Suzanne Hurtado at Suzanne.l.hurtado.civ@mail.mil, or (619) 607-1910.

Thanks!
Suzanne Hurtado
Principal Investigator
Evaluation of a Mobile Application for Prescription Drug Abuse Education (#NHRC.2016.0019)
Naval Health Research Center, San Diego, CA
(619) 607-1910, Email: Suzanne.l.hurtado.civ@mail.mil

#### 1-Month Survey Reminder Email

Dear study participant,

About one month ago you filled out a survey about the prevention of prescription medication misuse. Thanks for your participation! If you have already completed the 1-month survey for this study, thank you and please disregard this email. If you have not completed the 1-month survey, we now request that using a non-military mobile device or computer, you go to our study website: http://XXX and fill-out the 1-month survey for this study. Please submit it within the next three (3) days. The information you provide will be kept completely confidential.

As a thank you, when you submit this survey, you will receive \$25.00 in e-gift codes within approximately 2 business days. As a reminder, you must participate during off-duty, liberty or leave status if you wish to be compensated.

If you have any questions about the study, or if you do not wish to participate or be contacted any more, please contact Suzanne Hurtado at Suzanne.l.hurtado.civ@mail.mil, or (619) 607-1910.

Thanks!
Suzanne Hurtado
Principal Investigator
Evaluation of a Mobile Application for Prescription Drug Abuse Education (#NHRC.2016.0019)
Naval Health Research Center, San Diego, CA
(619) 607-1910, Email: Suzanne.l.hurtado.civ@mail.mil

APPROVED

DATE: 6 14 1/8

EXP: 6 1/4 1/9

Naval Health Research Center San Diego
#### 3-Month Survey Invitation Email

Dear study participant,

About two months ago you filled out a survey about the prevention of prescription medication misuse. Thanks for your participation! We now request that using a non-military mobile device or computer, you go to our study website: http://XXX and fill-out the 3-month survey for this study. Please submit it within the next three (3) days. The information you provide will be kept completely confidential.

As a thank you, when you submit this survey, you will receive \$50.00 in e-gift codes within approximately 2 business days. As a reminder, you must participate during off-duty, liberty or leave status if you wish to be compensated.

This is the last survey for this study. If you have any questions about the study, or if you do not wish to participate or be contacted any more, please contact Suzanne Hurtado at Suzanne.l.hurtado.civ@mail.mil, or (619) 607-1910.

Thanks!
Suzanne Hurtado
Principal Investigator
Evaluation of a Mobile Application for Prescription Drug Abuse Education (#NHRC.2016.0019)
Naval Health Research Center, San Diego, CA
(619) 607-1910, Email: Suzanne.l.hurtado.civ@mail.mil

#### 3-Month Survey Reminder Email

Dear study participant,

About two months ago you filled out a survey about the prevention of prescription medication misuse. Thanks for your participation! If you have already completed the 3-month survey for this study, thank you and please disregard this email. If you have not completed the 3-month survey, we now request that using a non-military mobile device or computer, you go to our study website: http://XXX and fill-out the 3-month survey for this study. Please submit it within the next three (3) days. The information you provide will be kept completely confidential.

As a thank you, when you submit this survey, you will receive \$50.00 in e-gift codes within approximately 2 business days. As a reminder, you must participate during off-duty, liberty or leave status if you wish to be compensated.

This is the last survey for this study. If you have any questions about the study, or if you do not wish to participate or be contacted any more, please contact Suzanne Hurtado at Suzanne.l.hurtado.civ@mail.mil, or (619) 607-1910.

Thanks!
Suzanne Hurtado
Principal Investigator
Evaluation of a Mobile Application for Prescription Drug Abuse Education (#NHRC.2016.0019)
Naval Health Research Center, San Diego, CA
(619) 607-1910, Email: Suzanne.l.hurtado.civ@mail.mil

DATE: 6 14 18 TD

EXP: 6 141 19

Naval Health Research Center San Diego

G. SURVEYS

Version Date: 14 MAY 2018

## [Online]

# Prescription Drug Awareness Survey

**Pretest** 

Naval Health Research Center 140 Sylvester Rd. San Diego, CA 92106-3521

APPROVED

DATE: 6 14 1/8

EXP: 6 1/4 1/9

Naval Health Research Center San Diego

## LOGIN

Please enter your non-DoD email address.

(Your email is the login for the surveys. This information will <u>not</u> be used for any other purpose. Once surveys are collected and linked together, your email address will be deleted from the study).

Your email address:

| | 100 |
|---|-----|
| A | |


APPROVED

DATE: 6 1 4 1 18

EXP: 6 1 4 1 79

Naval Health Research Center San Diego

| | DEMOGRAPHICS | | |
|---|---|---|---|
| 1. Are you male or female? | 5. What sexual orientation do you | 8. What is your | pay grade or rank? |
| O Male | consider yourself to be? | O E-1 | O Trainee |
| O Female | O Heterosexual | O E-2 | O W-1 to W-5 |
| | O Gay or lesbian | O E-3 | O O-1 or O-1E |
| 2. What is your ethnic background? | O Bisexual | O E-4 | O O-2 or O-2E |
| O Hispanic or Latino | O Other | O E-5 | O O-3 or O-3E |
| O Not Hispanic or Latino | O Don't Know | O E-6 | 0 0-4 |
| · | | O E-7 | O O-5 |
| 3. What is your race? | 6. How much education have you | O E-8 | O O-6 |
| O American Indian/Alaska Native | completed? | O E-9 | O-7 to O-10 |
| O Asian | O Did not complete high | | |
| O Native Hawaiian or Other | school or GED | 9. Have you eve | er been deployed? |
| Pacific Islander | O GED | O No O Y | · |
| O Black or African American | O Finished high school | | |
| O White | O Finished high school and | 10. How many | total combat |
| O Multi-racial | some college | deployments (ir | ncluding |
| O Other/unknown | O Associate's degree | peacekeeping n | nissions) have you |
| | O Bachelor's degree or higher | been on in your | military career? |
| 4. How old are you? | | O None | O 3 |
| (age) | 7. What is your Branch of service? | 01 | O 4 or more |
| , , , | O Navy | 0.2 | |
| | O Marine Corps | 02 | |
| | O Army | 550 | |
| | O Air Force | | |

## **MEDICATION AND PAIN**

O Coast Guard O Other: \_\_\_\_

## 11. Please answer the following.

| | No | Yes |
|---|---|---|
| a. Are you currently taking a prescription | medication? | 0 |
| b. Are you currently taking a prescription | PAIN medication? | 0 |
| c. Are you currently taking a prescription pain medication? | medication other than a O | 0 |




| | d. | Hurtado, Evaluation Are all your prescriptions filled through the same pl system? | | Abuse Educationa | ol App, Protocol | # NHRC. | 2016.0019<br>O |
|---|---|---|---|---|---|---|---|
| | | | | | No | Υ | 'es |
| | e. | Have you experienced an illness or injury for which currently being treated? | you are | | 0 | | 0 |
| | f. | Have you experienced an illness or injury for which experience chronic pain? | you still | | 0 | | 0 |
| YA | g. | Are you currently experiencing pain? | Sillo IS | | 0 | | 0 |
| | | TAKING MEDICATION | ON IN G | ENERAL | | | |
| 1 | 2. Pi | lease indicate how often the following has happene | ed to you | 1 | | | |
| | | | Never | Occasionally | Sometimes | Often | Always |
| | a. | At times I need to borrow pain medication from family and friends to get relief | 0 | 0 | 0 | 0 | 0 |
| | b. | I get pain medication from more than one doctor in order to have enough medication for my pain | 0 | 0 | 0 | 0 | 0 |
| | c. | At times I need to take medication more often than it is prescribed in order to relieve my pain | 0 | 0 | 0 | 0 | 0 |
| | d. | How many times in the <u>past year</u> have you asked your doctor to increase your prescribed dosage of pain medication in order to get relief? | 0 | 0 | 0 | 0 | 0 |
| | e. | How many times in the <u>past year</u> have you run out of pain medication early and had to request an early refill? | 0 | 0 | 0 | 0 | 0 |
| | f. | How many times in the <u>past year</u> have you accidentally misplaced your prescription for pain medication and had to ask for another? | 0 | 0 | 0 | 0 | 0 |
| | | MEDICATION LA | ST 30 D | AYS | | | |
| | | ease answer each question as honestly as possible<br>ganswers. If you are unsure about how to answer t | | | | | |
| | | (0) | Ne | ever Seldom | Sometimes | Often | Very<br>Often |
| | a. | In the past 30 days how often have you trouble with thinking clearly or had memory problems? | | 0 0 | 0 | 0 | 0 |
| | b. | In the past 30 days, how often do people complain | | 0 0 | 0 | 0 | 0 |
| V | ersion | Date: 14 MAY 2018 G-5 | | DATE | 1 | 8 10 | |

that you are not completing necessary tasks? (i.e., doing things that need to be done, such as going to class, work, or appointments)

| | | Never | Seldom | Sometimes | Often | very<br>Often |
|---|---|---|---|---|---|---|
| c. | In the past 30 days, how often have you had to go to someone other than your prescribing physician to get sufficient pain relief from medications? (i.e., another doctor, the Emergency Room, friends, street sources) | 0 | 0 | 0 | 0 | 0 |
| d. | In the past 30 days, how often have you taken your medications differently from how they are prescribed? | 0 | 0 | 0 | 0 | 0 |
| e. | thought about hurting yourself? | 0 | 0 | 0 | 0 | 0 |
| f. | In the past 30 days, how much of your time was spent thinking about opioid medications (having enough, taking them, dosing schedule, etc.)? | 0 | 0 | 0 | 0 | 0 |
| g. | In the past 30 days, how often have you been in an argument? | 0 | 0 | 0 | 0 | 0 |
| h. | In the past 30 days, how often have you had trouble controlling your anger (e.g., road rage, screaming, yelling, etc.)? | 0 | 0 | 0 | 0 | 0 |
| i. | In the past 30 days, how often have you needed to take pain medications belonging to someone else? | 0 | 0 | 0 | 0 | 0 |
| j. | In the past 30 days, how often have you been worried about how you're handling your medications? | 0 | 0 | 0 | 0 | 0 |
| k. | In the past 30 days, how often have others been worried about how you're handling your medications? | 0 | 0 | 0 | 0 | 0 |
| l. | In the past 30 days, how often have you had to make an emergency phone call or show up at the clinic without an appointment? | 0 | 0 | 0 | 0 | 0 |
| m. | In the past 30 days, how often have you gotten angry with people? | 0 | 0 | 0 | 0 | 0 |
| n. | In the past 30 days, how often have you had to take more of your medication than prescribed? | 0 | 0 | 0 | 0 | 0 |
| 0. | In the past 30 days, how often have you borrowed pain medication from someone else? | 0 | 0 | 0 | 0 | 0 |
| p. | In the past 30 days, how often have you used your pain medicine for symptoms other than for pain (e.g., to help you sleep, improve your mood, or relieve stress)? | 0 | O DATE: | APPROVED | 0 | °<br>] |
| Version | Date: 14 MAY 2018 G-6 | | EXP:<br>Naval H | 6 1141 19 | 2 J | |

| | Hurta q. In the past 30 days, how often have y the Emergency Room? | ado, Evaluation of a Dru<br>ou had to visit | O C | | Protocol # NHR O O | 27 27 27 27 2 |
|---|---|---|---|---|---|---|
| | | HOUSEHOLD | Tatolar Devi | | | |
| 1.4 | | HOUSEHOLD | | | | |
| 14. | Please answer the following. | | | | | |
| | The second secon | | | No | Υ | es |
| | Do you live with others? | | | 0 | | 0 |
| Ł | <ol> <li>Some types of medication pose a gr</li> </ol> | | 2. | 0 | ( | 0 |
| | These include some pain medications | • | | | | |
| | muscle relaxants, sleeping medication | · | • | | | |
| | medications among others. Is someor | • | d | | | |
| _ | or living quarters taking these types o | | | | | |
| • | Have you shared your prescription i | medication with | | 0 | | 0 |
| m. | others? | | | | es contract | |
| | | COMMUNICATIO | NI. | H 140 | | |
| | | COMMUNICATIO | | | | |
| <b>15.</b> | If you wanted to, how <u>prepared</u> do you | feel to talk to? | | | | |
| | | 3.4 m | | | | |
| | | Very | Somewhat | Neutral | Somewhat | Very |
| 2 | . Someone in your chain of command | unprepared | unprepared | | prepared | prepared |
| 2 | Someone in your <u>chain of command</u> if you were concerned about <u>YOUR</u> | 95999 | | Neutral<br>O | | • |
| a | | unprepared | unprepared | | prepared | prepared |
| a | if you were concerned about YOUR | unprepared | unprepared | | prepared | prepared |
| | if you were concerned about <u>YOUR</u> possible misuse of a prescribed | unprepared | unprepared | | prepared | prepared |
| | if you were concerned about YOUR possible misuse of a prescribed medication? | unprepared<br>O | unprepared<br>O | 0 | prepared<br>O | prepared |
| | if you were concerned about <u>YOUR</u> possible misuse of a prescribed medication? Your <u>doctor</u> if you were concerned | unprepared<br>O | unprepared<br>O | 0 | prepared<br>O | prepared |
| t | if you were concerned about <u>YOUR</u> possible misuse of a prescribed medication? Your <u>doctor</u> if you were concerned about <u>YOUR</u> possible misuse of a | unprepared<br>O | unprepared<br>O | 0 | prepared<br>O | prepared |
| t | if you were concerned about YOUR possible misuse of a prescribed medication? Your doctor if you were concerned about YOUR possible misuse of a prescribed medication? A buddy (fellow service member) if you were concerned about THEIR | unprepared<br>O | O O | 0 | prepared<br>O | o O |
| t | if you were concerned about YOUR possible misuse of a prescribed medication? Your doctor if you were concerned about YOUR possible misuse of a prescribed medication? A buddy (fellow service member) if you were concerned about THEIR possible misuse of a prescribed | unprepared<br>O | O O | 0 | prepared<br>O | o O |
| t | if you were concerned about YOUR possible misuse of a prescribed medication? Your doctor if you were concerned about YOUR possible misuse of a prescribed medication? A buddy (fellow service member) if you were concerned about THEIR possible misuse of a prescribed medication? | unprepared<br>O | O O | 0 | prepared<br>O | o<br>O |
| t | if you were concerned about YOUR possible misuse of a prescribed medication? Your doctor if you were concerned about YOUR possible misuse of a prescribed medication? A buddy (fellow service member) if you were concerned about THEIR possible misuse of a prescribed medication? A spouse (or significant other) if you | unprepared O O | O O | 0 | prepared<br>O | o<br>O |
| t | if you were concerned about YOUR possible misuse of a prescribed medication? Your doctor if you were concerned about YOUR possible misuse of a prescribed medication? A buddy (fellow service member) if you were concerned about THEIR possible misuse of a prescribed medication? A spouse (or significant other) if you were concerned about THEIR possible | unprepared O O | O O | 0 | prepared<br>O | prepared<br>O |
| t | if you were concerned about YOUR possible misuse of a prescribed medication? Your doctor if you were concerned about YOUR possible misuse of a prescribed medication? A buddy (fellow service member) if you were concerned about THEIR possible misuse of a prescribed medication? A spouse (or significant other) if you | unprepared O O | O O | 0 | prepared<br>O | prepared<br>O |
| t | if you were concerned about YOUR possible misuse of a prescribed medication? Your doctor if you were concerned about YOUR possible misuse of a prescribed medication? A buddy (fellow service member) if you were concerned about THEIR possible misuse of a prescribed medication? A spouse (or significant other) if you were concerned about THEIR possible | unprepared<br>O | O O | 0 | prepared<br>O | prepared<br>O |
| t d | if you were concerned about YOUR possible misuse of a prescribed medication? Your doctor if you were concerned about YOUR possible misuse of a prescribed medication? A buddy (fellow service member) if you were concerned about THEIR possible misuse of a prescribed medication? A spouse (or significant other) if you were concerned about THEIR possible misuse of a prescribed medication? | unprepared O ATTITUDES | O O | 0 | prepared<br>O | prepared<br>O |
| t d | if you were concerned about YOUR possible misuse of a prescribed medication? Your doctor if you were concerned about YOUR possible misuse of a prescribed medication? A buddy (fellow service member) if you were concerned about THEIR possible misuse of a prescribed medication? A spouse (or significant other) if you were concerned about THEIR possible | unprepared O ATTITUDES | O O | 0 | prepared<br>O | prepared<br>O |

G-7


Hurtado, Evaluation of a Drug Abuse Educational App, Protocol # NHRC.2016.0019

disagree agree nor agree

| | | GISUBICC | | disagree | | agree |
|---|---|---|---|---|---|---|
| a. | Misusing prescription drugs is dangerous. | 0 | 0 | 0 | 0 | 0 |
| | | Strongly<br>disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Strongly<br>agree |
| b. | Most service members misuse prescription drugs at some point while on active duty. | 0 | 0 | 0 | 0 | 0 |
| C. | It's not a big deal to share prescription medication with someone if you're trying to help them. | 0 | 0 | 0 | 0 | 0 |
| d. | It should be illegal to share prescription medication with friends. | 0 | 0 | 0 | 0 | 0 |
| e. | It should be illegal to share prescription medication with family members. | 0 | 0 | 0 | 0 | 0 |
| f. | If you've been prescribed medication by your doctor, you should take it only as directed. | 0 | 0 | 0 | 0 | 0 |
| g. | If you share your prescription medications with friends or family, you are putting their health at risk. | 0 | 0 | 0 | 0 | 0 |
| h. | The risk of getting in trouble for taking pain medication differently than prescribed is a concern for me. | 0 | 0 | 0 | 0 | 0 |
| i. | There is a high risk of getting caught if you take your own old prescription medication. | 0 | 0 | 0 | 0 | 0 |
| j. | Using someone else's prescription medication can be hazardous to your health. | 0 | 0 | 0 | 0 | 0 |
| k. | Using someone else's prescription medication can cost you your military career. | 0 | 0 | 0 | 0 | 0 |
| l. | It is no big deal if I take a higher dose of my prescription pain reliever than directed. | 0 | 0 | 0 | 0 | 0 |
| | It is risky to my health to take my medication more often than prescribed. | 0 | 0 | 0 | 0 | 0 |
| n. | Even if a medication label says not to take it with alcohol, it is ok to take it with only one drink. | 0 | 0 | 0 | 0 | 0 |
| 0. | is only risky if you are binge drinking. | rs O | 0 | 0 | 0 | 0 |
| | If I have questions about a prescription Date: 14 MAY 2018 | O<br>G-8 | DAT | O<br>APPROV<br>E: 6 / 4 | | P |

| | | Strongly<br>disagree | Disagree | Neither agree nor disagree | Agree | Strongly<br>agree |
|---|---|---|---|---|---|---|
| r. | If is important to read the label on my prescription medication. | 0 | 0 | 0 | 0 | 0 |
| S. | It is important to read the material that the pharmacy provides with my prescription medication. | 0 | 0 | 0 | 0 | 0 |
| t. | If I have concerns about my medication, it's important that I know where to go for information. | 0 | 0 | 0 | 0 | 0 |
| u. | It is ok to use your leftover prescription medication for a new condition. | 0 | 0 | 0 | 0 | 0 |
| v. | There is nothing wrong with taking an extra dose of my prescription pain reliever if I am in pain. | 0 | 0 | 0 | 0 | 0 |

## 17. Please indicate how much you agree or disagree with the statements.


| | | Strongly<br>disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Strongly<br>agree |
|---|---|---|---|---|---|---|
| a. | There are certain situations where it is ok | 0 | 0 | 0 | 0 | 0 |
| | to take someone else's prescribed medication. | | | | | |
| b. | If a person is in physical pain from an injury, taking someone else's prescription medication is okay. | 0 | 0 | 0 | 0 | 0 |
| C. | As long as it makes you feel better and not worse, it's fine to take prescription drugs while drinking. | 0 | 0 | 0 | 0 | 0 |
| d. | An individual should only take medication that is prescribed to them by a medical professional. | 0 | 0 | 0 | 0 | 0 |
| e. | It is acceptable | 0 | ОГ | U ADDD | Overs | -01 |

G-9

Hurtado, Evaluation of a Drug Abuse Educational App, Protocol # NHRC.2016.0019 for a fellow service member to borrow someone's prescription medication in order to enhance their readiness. f. It is ok for a 0 0 0 0 0 service member to take medication that is not prescribed to them in order to decrease appetite and lose weight. Strongly Disagree Neither Agree Strongly disagree agree nor agree disagree Using prescribed g. 0 0 0 0 0 medications to stay awake for duty is okay. h. Taking 0 0 0 0 0 medication that is not prescribed to you should be illegal. 18. How much do you think people <u>risk harming themselves</u> (physically or in other ways) by...?

| | | | No risk | Slight risk | Moderate<br>risk | Great risk |
|---|---|---|---|---|---|---|
| a. | prescription drug<br>(examples: oxycodone, Valiu | Taking <u>someone else's</u> m)? | 0 | 0 | 0 | 0 |
| b. | (examples: oxycodone,<br>Valium) in <u>higher doses</u> than | Taking prescription drug what a doctor prescribed? | 0 | 0 | 0 | 0 |
| c. | drug (examples: oxycodone, Valium) together with alcohol | Taking a prescription ol or other drugs? | 0 | 0 | 0 | 0 |
| d. | of alcohol once or twice each weekend? | Having <u>5 or more drinks</u> | 0 | 0 | 0 | 0 |
| e. | regularly (more than once a week)? | Smoking <u>marijuana</u> | 0 | 0 | 0 | 0 |

#### 19. Please indicate how much you agree or disagree with the statements.

Strong y Disagraphroven Strongly

DATE: 6 14 18 10

EXP: 6 117 19


G-10

| | 2.72 | | disagree | | | agree |
|---|---|---|---|---|---|---|
| a. | to stay away from misusing prescription drugs oxycodone, Valium). | I have made a final decision (examples: | 0 | 0 | 0 | 0 |
| b | to stay away from | I have made a final decision (examples: oxycodone, Valium). | 0 | 0 | 0 | Ö |
| C. | prescription medications exactly as prescribed by my | I intend to use my provider. | 0 | 0 | 0 | 0 |
| d. | someone misusing prescription medication. | I plan to intervene if I see | 0 | 0 | 0 | 0 |

Please continue onto next page.

#### **KNOWLEDGE**

- 20. Based upon DoD policy, which of the following is NOT an example of prescription drug misuse?
  - a. Taking more of your medication that is prescribed
  - b. Taking your medication at 2150 instead of 2200 because you plan to go to sleep
  - c. Using the prescription you got earlier this year for your knee for a back strain you got this week
  - d. Taking your pain medication 4 times a day instead of 3 like it says on the label
  - e. Giving some of your medication to your spouse because he or she ran out
- **21.** Which of the following is <u>NOT</u> a recommendation in the Prescription for Discharge campaign to protect Sailors and Marines from prescription drug misuse/abuse?
  - a. Report promptly
  - b. Take correctly
  - c. Save for emergencies
  - d. Never share
  - e. Dispose properly
- **22.** What should a service member do if they receive a prescription medication from a *non-military* medical treatment facility?

G-11

a. Report it to the Chaplain


APPROVED

DATE: 6 / 4 / /8

EXP: 6 / 14 / 19

Naval Health Research Center San Diego

- b. It ONLY needs to be reported to their military health care provider if they had an adverse reaction
- c. It does not need to be reported
- d. Report it to their military health care provider at their next visit
- e. Report it to their chain of command and ensure it is entered into their military health record
- 23. What type of alternative treatment involves visualizing specific positive scenes to reduce stress?
  - a. Biofeedback
  - b. Acupuncture
  - c. Yoga
  - d. Guided Imagery
  - e. Physical Therapy
- **24.** What type of alternative treatment involves becoming mindful of one's thoughts and sensations in a nonjudgmental way?
  - a. Physical Therapy
  - b. Biofeedback
  - c. Chiropractic Therapies
  - d. Massage Therapy
  - e. Meditation
- 25. What can you do if you suspect someone is misusing prescription medication?
  - a. Provide support
  - b. Be a role model
  - c. Keep medications safe and secured
  - d. Inform chain of command or law enforcement officials
  - e. All of the above
- 26. Which of the following is NOT potentially a sign or symptom associated with prescription drug misuse?
  - a. Relationship problems
  - b. Sudden weight loss or gain
  - c. Asking your doctor questions about your prescription
  - d. Changes in appetite or sleep patterns
  - e. Decreased performance at work
- 27. What are the two most commonly misused prescription drugs among military personnel?
  - a. Pain relievers (opioids) and central nervous system depressants (sedatives
  - b. Pain relievers (opioids) and protease inhibitors
  - c. Central nervous system depressants (sedatives) and protease inhibitors
  - d. Central nervous system depressants (sedatives) and central nervous system stimulants

G-12

e. Pain relievers (opioids) and central nervous system stimulants

APPROVED

DATE: 6 | 4 | 18

EXP: 6 | 14 | 19

Naval Health Research Center San Diego


- 28. Which of the following is a negative consequence of misusing prescription drugs?
  - a. Drug addiction
  - b. Altered judgment
  - c. Unintentional overdose
  - d. Drug tolerance
  - e. All of the above
- 29. What is a specific sign or symptom of prescription drug misuse?
  - a. Faking illness or injury to obtain medications
  - b. Excessive visits to the doctor
  - c. Stealing, forging, or selling prescriptions
  - d. None of the above
  - e. All of the above
- 30. Which of the following could help you reduce your risk of prescription drug misuse? (Select the best answer)
  - a. Ask your friend which medication worked best for them to treat pain
  - b. Take your old prescription for pain without consulting your doctor
  - c. Wait until your pain is unbearable before taking pain medication instead of taking it at the regular intervals indicated
  - d. Talk to your doctor about symptoms you may be having or concerns about your medication
  - e. Mix your prescription medication with over-the-counter medicine and supplements
- **31.** It is important to talk to your doctor or pharmacist about ... (Select the best answer)
  - a. Using over-the-counter medications while using your prescription
  - b. Supplements that you routinely take
  - c. Symptoms and side effects you are experiencing
  - d. A and C
  - e. All of the above
- 32. TRUE OR FALSE: Everyday activities such as playing sports cannot cause traumatic brain injuries (TBI).
  - a. TRUE
  - b. FALSE
- 33. TRUE OR FALSE: Prescription drugs are regulated so they are always safe to take.
  - a. TRUE
  - b. FALSE
- 34. TRUE or FALSE: It is safe to take prescription medication from a previous health problem to treat new symptoms.

a. TRUE

Version Date: 14 MAY 2018 G-13

APPROVED

DATE: 6 1 4 1 18

EXP: 6 1 4 1 9

Navel Health Research Center San Diego

- **35.** Which of the following is a good resource for someone seeking information about a prescription medication misuse problem? (Select all that apply)
  - a. SACO or DAPA
  - b. Corpsman or other medical provider
  - c. Commanding Officer
  - d. Diversity Officer
  - e. MilitaryOneSource
- 36. Drinking alcohol with prescription medication can do which of the following? (Select all that apply)
  - a. Increase side effects
  - b. Increase effectiveness
  - c. Decrease effectiveness
  - d. Decrease sedative effects
  - e. Increase risk of a toxic reaction
- **37.** Which of the following has contributed to the increase in prescription drug abuse among service members? (Select all that apply)
  - a. Increase in prescriptions for pain related to injuries among OIF and OEF veterans
  - b. Decrease in military pharmacy regulations
  - c. Increase in average working hours among service members
  - d. Decrease in the number of compounds tested in drug screening
  - e. Increase in the number of military health care providers
- 38. Which step(s) can you take to reduce prescription drug misuse? (Select all that apply)
  - a. Use previously prescribed medication for a current health issue
  - b. Keep your medications safe and secured
  - c. Only borrow prescription medication from a spouse or other trusted source
  - d. Dispose of unused or expired prescription medication properly
  - e. Do not share medication
- **39.** Which of the following are key points you would want to discuss with your pharmacist when getting a new prescription? (Select all that apply)
  - a. Best time of day to take medication
  - b. Other health conditions the medications may be used for in the future
  - c. Prescribed dosage
  - d. Potential side effects and warnings
  - e. Alternative non-medical treatments

**40.** Which of the following are signs and symptoms of depression? (Select all that apply Version Date: 14 MAY 2018 G-14



- a. Changes in appetite or weight
- b. Increased motivation
- c. Increased energy
- d. Decreased energy
- e. Irritability
- **41.** Which of the following statement(s) about sleep is TRUE? (Select all that apply)
  - a. The quality of sleep you are getting is just as important as the amount
  - b. Sleep problems can be a side effect of some medications
  - c. The amount of sleep you are getting is the most important aspect of sleep
  - d. Sleep problems can be a symptom of a mental health condition
  - e. Catching-up on sleep is just as effective as regular sleep
- 42. What are two common forms of treatment for mental health conditions such as depression, anxiety, and PTSD? (Select all that apply)
  - a. Medication
  - b. Physical therapy
  - c. Dietary changes
  - d. No treatment available
  - e. Psychotherapy

#### STRESS AND HISTORY

## 43. Over the last 2 weeks, how often have you been bothered by the following problems?

| | | Not at all | Several days | More than half the days | Nearly<br>every day |
|---|---|---|---|---|---|
| a. | Feeling nervous, anxious or on edge | 0 | 0 | 0 | 0 |
| b. | Not being able to stop or control worrying | 0 | 0 | 0 | 0 |
| c. | Feeling down, depressed, or hopeless | 0 | 0 | 0 | 0 |
| d. | Little interest or pleasure in doing things | 0 | 0 | 0 | 0 . |

#### 44. Have you ever had any experience that was so frightening, horrible, or upsetting that, IN THE PAST MONTH, you...

| | No | Yes | |
|---|---|---|---|
| a. Have had nightmares about it or thought about it when | 0 | 0 | |
| you did not want to? | | | 1 |
| b. Tried hard not to think about it or went out of your way | 0 | 0 | |
| to avoid situations that remind you of it? | | | |
| c. Were constantly on guard, watchful, or easily startled? | 0 | 0 | 1 |
| d. Felt numb or detached from others, activities, or | ØATE: 6 | 4 1/8 0 | 4 |
| Version Date: 14 MAY 2018 G-15 | EXP: 6 11 | 4119 70 | |

Naval Health Research Center San Diego

| | No | Yes |
|---|---|---|
| 45. Have you ever been on a deployment where you felt | 0 | 0 |
| you were in imminent danger? | | |
| 46. If "yes" to above, did you have any injury(ies) during your deplall that apply). | oyment from a | ny of the following? (Mar |
| O Fragment | | |
| O Bullet | | |
| O Vehicular | | 22 |
| O Fall | | |
| O Blast (Improvised explosive device, RPG, land mine, grenad | e, etc.) | |
| O Other | | |
| Please continue onto next | page. | |
| 47. Did any injury received while you were deployed result in any | of the following | ng? (Mark all that apply). |
| O Being dazed, confused or "seeing stars" | | |
| O Not remembering the injury | | |
| O Losing consciousness (knocked out) for less than a minute | | |
| O Losing consciousness for 1-20 minutes | | |
| O Losing consciousness for longer than 20 minutes | | = |
| O Having symptoms of concussion afterward (such as headac | he, dizziness, ir | ritability, etc.) |
| O Head injury | | |
| O None of the above | | |
| 48. Have you ever had a problem with substance abuse? | No 🔿 | Yes O |
| CLIDAAT CLIDVEV | | |

SUBMIT SURVEY

Thanks for completing this survey! We greatly appreciate your participation!

G-16


APPROVED

DATE: 6 1 4 1 18

EXP: 6 114 1 19 JD

Naval Health Research Center San Diego

## [Online]

# Prescription Drug Awareness Survey

1-month posttest (intervention group)

Protocol # NHRC.2016.0019

Naval Health Research Center

140 Sylvester Rd.

San Diego, CA 92106-3521

APPROVED

DATE: 6 | 4 | 18

EXP: 6 | 14 | 19

Navai Health Research Center San Diego

#### LOGIN

Please enter your non-DoD email address.

(Your email is the login for the surveys. This information will <u>not</u> be used for any other purpose. Once surveys are collected and linked together, your email address will be deleted from the study.)

Your E-mail address:

DATE: 6 14 1/8
EXP: 6 1/4 1/9
Naval Health Research Center San Diego

#### **MEDICATION AND PAIN**

## 1. Please answer the following.

| | | No | Yes |
|---|---|---|---|
| a. | Are you currently taking a prescription medication? | 0 | 0 |
| b. | Are you currently taking a prescription PAIN medication? | 0 | 0 |
| C. | Are you currently taking a prescription medication other than a pain medication? | 0 | 0 |
| d. | Are all of your prescriptions filled through the same pharmacy system? | 0 | 0 |
| e. | Have you experienced an illness or injury for which you are currently being treated? | 0 | 0 |
| f. | Have you experienced an illness or injury for which you still experience chronic pain? | 0 | 0 |
| g. | Are you currently experiencing pain? | 0 | 0 |

#### **TAKING MEDICATION IN GENERAL**

#### 2. Please indicate how often the following has happened to you...

| | | Never | Occasionally | Sometimes | Often | Always |
|---|---|---|---|---|---|---|
| a. | At times I need to borrow pain medication from friends or family to get relief | 0 | 0 | 0 | 0 | 0 |
| b. | I get pain medication from more than one doctor in order to have enough medication for my pain | 0 | 0 | 0 | 0 | 0 |
| C. | At times I need to take medication more often than it is prescribed in order to relieve my pain | 0 | 0 | 0 | 0 | 0 |
| d. | How many times in the <u>past year</u> have you asked your doctor to increase your prescribed dosage of pain medication in order to get relief? | 0 | 0 | 0 | 0 | 0 |
| e. | How many times in the <u>past year</u> have you run out of pain medication early and had to request an early refill? | 0 | 0 | 0 | 0 | 0 |
| f. | How many times in the <u>past year</u> have you accidentally misplaced your prescription for pain medication and | 0 | 0 | 0 | 0 | 0 |
| | had to ask for another? | | | | APPROVED | - |

DATE: 6 14 1/8
EXP: 6 141 19
Naval Health Research Center San Diego

#### **MEDICATION LAST 30 DAYS**

3. Please answer each question as honestly as possible regarding the <u>past 30 days</u>. There are no right or wrong answers. If you are unsure about how to answer the question, please give the best answer you can.

| answer you can. | | | | | |
|---|---|---|---|---|---|
| | Never | Seldom | Sometimes | Often | Very<br>often |
| a. In the past 30 days, how often have you had trouble with thinking clearly or had memory problems? | 0 | 0 | 0 | 0 | 0 |
| b. In the past 30 days, how often do people<br>complain that you are not completing<br>necessary tasks? (i.e., doing things that<br>need to be done, such as going to class,<br>work or appointments) | 0 | 0 | 0 | 0 | 0 |
| c. In the past 30 days, how often have you had to go to someone other than your prescribing physician to get sufficient pain relief from medications? (i.e., another doctor, the Emergency Room, friends, street sources) | 0 | 0 | 0 | 0 | 0 |
| d. In the past 30 days, how often have you<br>taken your medications differently from<br>how they are prescribed? | 0 | 0 | 0 | 0 | 0 |
| e. In the past 30 days, how often have you seriously thought about hurting yourself? | 0 | 0 | 0 | 0 | 0 |
| f. In the past 30 days, how much of your<br>time was spent thinking about opioid<br>medications (having enough, taking<br>them, dosing schedule, etc.)? | 0 | 0 | 0 | 0 | 0 |
| g. In the past 30 days, how often have you been in an argument? | 0 | 0 | 0 | 0 | 0 |
| h. In the past 30 days, how often have you<br>had trouble controlling your anger (e.g.,<br>road rage, screaming, yelling, etc.)? | 0 | 0 | 0 | 0 | 0 |
| i. In the past 30 days, how often have you needed to take pain medications belonging to someone else? | 0 | 0 | 0 | 0 | 0 |
| j. In the past 30 days, how often have you been worried about how you're handling your medications? | 0 | 0 | DATE: 6 / EXP: 6 / Naval Health Res | PROVED 4 1/8 14 1/9 earch Center San | Diego |
| 0.00 | G-20 | | | | |

G-20

| | | Never | Seldom | Sometimes | Often | Very<br>often |
|---|---|---|---|---|---|---|
| k. | In the past 30 days, how often have others been worried about how you're handling your medications? | 0 | 0 | 0 | 0 | 0 |
| I. | In the past 30 days, how often have you had to make an emergency phone call or show up at the clinic without an appointment? | 0 | 0 | 0 | 0 | 0 |
| m. | In the past 30 days, how often have you gotten angry with people? | 0 | 0 | 0 | 0 | 0 |
| n. | In the past 30 days, how often have you had to take more of your medication than prescribed? | 0 | 0 | 0 | 0 | 0 |
| 0. | In the past 30 days, how often have you borrowed pain medication from someone else? | 0 | 0 | 0 | 0 | 0 |
| p. | In the past 30 days, how often have you used your pain medicine for symptoms other than for pain (e.g., to help you sleep, improve your mood, or relieve stress)? | 0 | 0 | 0 | 0 | 0 |
| q. | In the past 30 days, how often have you had to visit the Emergency Room? | 0 | 0 | 0 | 0 | 0 |

#### HOUSEHOLD

## 4. Please answer the following.

| | | No | Yes | |
|---|---|---|---|---|
| a. | Do you live with others? | 0 | 0 | |
| b. | Some types of medication pose a greater risk of misuse. These include some pain medications, benzodiazepines muscle relaxants, sleeping medications, and some anxiety medications among others. Is someone in your household or living quarters taking these types of medications? | 0 | 0 | |
| c. | Have you shared your prescription medication with others? | 0 | 0 | . vector |

Please continue onto next page.

APPROVED

DATE: 6 1 4 1 18

EXP: 6 1 4 1 19

Naval Health Research Center San Diego

#### COMMUNICATION 5. If you wanted to, how prepared do Very Somewhat Somewhat Very unprepared prepared unprepared Neutral prepared you feel to talk to ...? a. Someone in your chain of command 0 0 0 0 0 if you were concerned about YOUR possible misuse of a prescribed medication? b. Your doctor if you were concerned 0 0 0 0 0 about YOUR possible misuse of a prescribed medication? c. A buddy (fellow service member) if 0 0 0 0 0 you were concerned about THEIR possible misuse of a prescribed medication? d. A spouse (or significant other) if you 0 0 0 0 0 were concerned about THEIR possible misuse of a prescribed medication? **ATTITUDES**

#### 6. Please indicate how much you agree or disagree with the statements.

| | | Strongly<br>disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Strongly<br>agree |
|---|---|---|---|---|---|---|
| a. | Misusing prescription drugs is dangerous. | 0 | 0 | 0 | 0 | 0 |
| b. | Most service members misuse prescription drugs at some point while on active duty. | 0 | 0 | 0 | 0 | 0 |
| c. | It's not a big deal to share prescription medication with someone if you're trying to help them. | 0 | 0 | 0 | 0 | 0 |
| d. | It should be illegal to share prescription medication with friends. | 0 | 0 | 0 | 0 | 0 |
| e. | It should be illegal to share prescription medication with family members. | 0 | 0 | 0 | 0 | 0 |
| f. | If you've been prescribed medication by your doctor, you should take it only as directed. | 0 | 0 | 0 | 0 | 0 |
| g. | If you share your prescription medications with friends or family, you are putting their health at risk. | 0 | 0 | 0 | 0 | 0 |
| | | Strongly<br>disagree | Disagree | Neither<br>agree nor | Agree<br>APPROVED | agree |

agree nor disagree disagree & 14/18 TLD

EXP: 6/14/19 TLD

Naval Health Research Center San Diego

G-22

| - | The risk of getting in trouble for taking pain medication differently than prescribed is a concern for me. | 0 | 0 | 0 | 0 | 0 |
|---|---|---|---|---|---|---|
| i. | There is a high risk of getting caught if you take your own old prescription medication. | 0 | 0 | 0 | 0 | 0 |
| j. | Using someone else's prescription medication can be hazardous to your health. | 0 | 0 | 0 | 0 | 0 |
| k. | Using someone else's prescription medication can cost you your military career. | 0 | 0 | 0 | 0 | 0 |
| 1. | It is no big deal if I take a higher dose of my prescription pain reliever than directed. | 0 | 0 | 0 | 0 | 0 |
| m. | It is risky to my health to take my medication more often than prescribed. | 0 | 0 | 0 | 0 | 0 |
| n. | Even if a medication label says not to take it with alcohol, it is ok to take it with only one drink. | 0 | 0 | 0 | 0 | 0 |
| 0. | Drinking alcohol with prescription pain relievers is only risky if you are binge drinking. | 0 | 0 | 0 | 0 | 0 |
| p. | If I have questions about a prescription medication, I should ask my provider. | 0 | 0 | 0 | 0 | 0 |
| | If I have questions about a prescription medication, I should ask the pharmacy tech. | 0 | 0 | 0 | 0 | 0 |
| r. | It is important to read the label on my prescription medication. | 0 | 0 | 0 | 0 | 0 |
| s. | It is important to read the material that the pharmacy provides with my prescription medication. | 0 | 0 | 0 | 0 | 0 |
| t. | If I have concerns about my medication, it's important that I know where to go for information. | 0 | 0 | 0 | 0 | 0 |
| u. | It is ok to use your leftover prescription medication for a new condition. | 0 | 0 | 0 | 0 | 0 |
| v. | There is nothing wrong with taking an extra dose of my prescription pain reliever if I am in pain. | 0 | 0 | 0 | 0 | 0 |

7. Please indicate how much you agree or disagree with the statements.

APPROVED

DATE: 6 1 4 1 18

EXP: 6 1 14 1 19

Naval Health Research Center San Diego

| | Hundo, Evaluati | - | | 732 T T | # 14111C.201 | 0.0017 |
|---|---|---|---|---|---|---|
| | | Strongly<br>disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Strongly<br>agree |
| a. | There are certain situations where it is ok to take someone else's prescribed medication. | 0 | 0 | 0 | 0 | 0 |
| b. | If a person is in physical pain from an injury, taking someone else's prescription medication is okay. | 0 | 0 | 0 | 0 | 0 |
| C. | As long as it makes you feel better and not worse, it's fine to take prescription drugs while drinking. | 0 | 0 | 0 | 0 | 0 |
| d. | An individual should only take medication that is prescribed to them by a medical professional. | 0 | 0 | 0 | 0 | 0 |
| e. | It is acceptable for a fellow service member to borrow someone's prescription medication in order to enhance their readiness. | 0 | 0 | 0 | 0 | 0 |
| f. | It is ok for a service member to take medication that is not prescribed to them in order to decrease appetite and lose weight. | 0 | 0 | 0 | 0 | 0 |
| g. | Using prescribed medications to stay awake for duty is okay. | 0 | 0 | 0 | 0 | 0 |
| h. | Taking medication that is not prescribed to you should be illegal. | 0 | 0 | 0 | 0 | 0 |

## 8. How much do you think people <u>risk harming themselves</u> (physically or in other ways) by...?

| | No risk | Slight risk | Moderate<br>risk | Great risk |
|---|---|---|---|---|
| a. Taking <u>someone else's</u> prescription drug (examples: oxycodone, Valium)? | 0 | 0 | 0 | 0 |
| b. Taking a prescription drug (examples: oxycodone,<br>Valium) in <u>higher doses</u> than what a doctor<br>prescribed? | 0 | 0 | 0 | 0 |
| c. Taking a prescription drug (examples: oxycodone, Valium) together with alcohol or other drugs? | 0 | DATE: EXP: Naval H | APPROVED 6 1411 6 11411 ealth Research Cent | 8 JLO<br>g San Diego |

| Hurtado, Evaluation of a D | Hurtado, Evaluation of a Drug Abuse Educational App, Protocol # NHRC.2016.0019 | | | |
|---|---|---|---|---|
| d. Having 5 or more drinks of alcohol once or twice<br>each weekend? | 0 | 0 | 0 | 0 |
| e. Smoking marijuana regularly (more than once a week)? | 0 | 0 | 0 | 0 |
| 9. Please indicate how much you agree or disagree | with the stat | ements. | | |
| | Strongly<br>disagree | Disagree | Agree | Strongly agree |
| a. I have made a final decision to stay away from<br>misusing prescription drugs (examples:<br>oxycodone, Valium). | 0 | 0 | 0 | 0 |
| b. I have made a final decision to stay away from<br>abusing prescription drugs (examples: oxycodone,<br>Valium). | 0 | 0 | 0 | 0 |
| c. I intend to use my prescription medications exactly as prescribed by my provider. | 0 | 0 | 0 | 0 |
| d. I plan to intervene if I see someone misusing prescription medication. | 0 | 0 | 0 | 0 |
| KNOWLE | DGE | | | |
| <ul> <li>10. Based upon DoD policy, which of the following is NO a. Taking more of your medication that is prescribed b. Taking your medication at 2150 instead of 2200 because. Using the prescription you got earlier this year for your d. Taking your pain medication 4 times a day instead of 3 e. Giving some of your medication to your spouse because</li> <li>11. Which of the following is NOT a recommendation in protect Sailors and Marines from prescription drug in a. Report promptly b. Take correctly c. Save for emergencies d. Never share e. Dispose properly</li> <li>12. What should a service member do if they receive a patreatment facility?</li> </ul> | se you plan to<br>r knee for a ba<br>like it says on<br>se he or she rai<br>n the Prescripti<br>nisuse/abuse? | go to sleep<br>ck strain you go<br>the label<br>n out<br>ion for Discharg | ot this week | to |
| a. Report it to the Chaplain b.It ONLY needs to be reported to their military health ca | are provider if | they had an ad | verse reactio<br>APPROV | VED. |
| c. It does not need to be reported d. Report it to their military health care provider at their i | next visit | DAT<br>EXI<br>Nava | E: <u>6 14</u><br>P: <u>6 114</u><br>I Health Research | 1/8 JD<br>1/9 Center San Diego |

G-25

Vomine Date: 14 MAY 2019

- e.Report it to their chain of command and ensure it is entered into their military health record
- 13. What type of alternative treatment involves visualizing specific positive scenes to reduce stress?
- a. Biofeedback
- b.Acupuncture
- c. Yoga
- d.Guided Imagery
- e. Physical Therapy
- 14. What type of alternative treatment involves becoming mindful of one's thoughts and sensations in a nonjudgmental way?
- a. Physical Therapy
- b.Biofeedback
- c. Chiropractic Therapies
- d. Massage Therapy
- e.Meditation
- 15. What can you do if you suspect someone is misusing prescription medication?
- a. Provide support
- b.Be a role model
- c. Keep medications safe and secured
- d.Inform chain of command or law enforcement officials
- e.All of the above
- 16. Which of the following is NOT potentially a sign or symptom associated with prescription drug misuse?
  - a. Relationship problems
  - b.Sudden weight loss or gain
  - c. Asking your doctor questions about your prescription
  - d. Changes in appetite or sleep patterns
  - e. Decreased performance at work
- 17. What are the two most commonly misused prescription drugs among military personnel?
  - a. Pain relievers (opioids) and central nervous system depressants (sedatives)
  - b. Pain relievers (opioids) and protease inhibitors
  - c. Central nervous system depressants (sedatives) and protease inhibitors
  - d.Central nervous system depressants (sedatives) and central nervous system stimulants
    Pain relievers (opioids) and central nervous system stimulants
- 18. Which of the following is a negative consequence of misusing prescription drugs?
  - a. Drug addiction
  - b.Altered judgment
  - c. Unintentional overdose
  - d.Drug tolerance
  - e.All of the above
- 19. What is a specific sign or symptom of prescription drug misuse?
  - a. Faking illness or injury to obtain medications
  - b. Excessive visits to the doctor
  - c. Stealing, forging, or selling prescriptions
  - d. None of the above



#### e.All of the above

- 20. Which of the following could help you reduce your risk of prescription drug misuse? (Select the best answer)
  - a. Ask your friend which medication worked best for them to treat pain
  - b. Take your old prescription for pain without consulting your doctor
  - c. Wait until your pain is unbearable before taking pain medication instead of taking it at the regular intervals indicated
  - d. Talk to your doctor about symptoms you may be having or concerns about your medication
  - e.Mix your prescription medication with over-the-counter medicine and supplements
- 21. It is important to talk to your doctor or pharmacist about... (Select the best answer)
  - a. Using over-the-counter medications while using your prescription
  - b. Supplements that you routinely take
  - c. Symptoms and side effects you are experiencing
  - d.A and C
  - e.All of the above
- 22. TRUE OR FALSE: Everyday activities such as playing sports cannot cause traumatic brain injuries (TBI).
  - a.TRUE
  - **b.FALSE**
- 23. TRUE OR FALSE: Prescription drugs are regulated so they are always safe to take.
  - a.TRUE
  - b.FALSE
- 24. TRUE OR FALSE: It is safe to take prescription medication from a previous health problem to treat new symptoms.
  - a.TRUE
  - **b.FALSE**
- 25. Which of the following is a good resource for someone seeking information about a prescription medication misuse problem? (Select all that apply)
- a. SACO or DAPA
- b.Corpsman or other medical provider
- c. Commanding Officer
- d.Diversity Officer
- e.MilitaryOneSource
- 26. Drinking alcohol with prescription medication can do which of the following? (Select all that apply)
  - a. Increase side effects
  - b.Increase effectiveness
  - c. Decrease effectiveness
  - d.Decrease sedative effects
  - e. Increase risk of a toxic reaction

DATE: 6 1/1/18
EXP: 6 1/4/19
Naval Health Research Center San Diego

- 27. Which of the following has contributed to the increase in prescription drug abuse among service members? (Select all that apply)
  - a. Increase in prescriptions for pain related to injuries among OIF and OEF veterans
  - b. Decrease in military pharmacy regulations
  - c. Increase in average working hours among service members
  - d.Decrease in the number of compounds tested in drug screening
  - e.Increase in the number of military health care providers
- 28. Which step(s) can you take to reduce prescription drug misuse? (Select all that apply)
  - a. Use previously prescribed medication for a current health issue
  - b. Keep your medications safe and secured
  - c. Only borrow prescription medication from a spouse or other trusted source
  - d. Dispose of unused or expired prescription medication properly
  - e.Do not share medication
- 29. Which of the following are key points you would want to discuss with your pharmacist when getting a new prescription? (Select all that apply)
  - a. Best time of day to take medication
  - b.Other health conditions the medication may be used for in the future
  - c. Prescribed dosage
  - d.Potential side effects and warnings
  - e. Alternative non-medical treatments
- 30. Which of the following are signs and symptoms of depression? (Select all that apply)
  - a. Changes in appetite or weight
  - b.Increased motivation
  - c. Increased energy
  - d.Decreased energy
  - e.Irritability
- **31.** Which of the following statement(s) about sleep is TRUE? (Select all that apply)
  - a. The quality of sleep you are getting is just as important as the amount
  - b. Sleep problems can be a side effect of some medications
  - c. The amount of sleep you are getting is the most important aspect of sleep
  - d.Sleep problems can be a symptom of a mental health condition
  - e. Catching-up on sleep is just as effective as regular sleep
- **32.**What are two common forms of treatment for mental health conditions such as depression, anxiety, and PTSD? (Select all that apply)
  - a. Medication
  - b. Physical therapy
  - c. Dietary changes
  - d.No treatment available
  - e. Psychotherapy

DATE: 6 14 118 DE Naval Health Research Center San Diego

#### **RATINGS OF THE APP**

## 33. Please rate the various aspects of the app.

| | W | Disliked<br>very much | Disliked | Neither<br>liked nor<br>disliked | Liked | Liked very<br>much |
|---|---|---|---|---|---|---|
| a. | The app as a whole | 0 | 0 | 0 | 0 | 0 |
| b. | Overall content | 0 | 0 | 0 | 0 | 0 |
| c. | Overall appearance and graphics | 0 | 0 | 0 | 0 | 0 |

34. Please indicate how much you agree or disagree with the statements.

| 34. Please indicate now much you agree or d | isagree with | tne stateme | nts. | | |
|---|---|---|---|---|---|
| | Strongly<br>disagree | Disagree | Neither agree nor disagree | Agree | Strongly<br>agree |
| a. The app was <u>useful</u> | 0 | 0 | 0 | 0 | 0 |
| <b>b.</b> I learned <u>new</u> information from this app | 0 | 0 | 0 | 0 | 0 |
| c. The app was <u>easy</u> to use | 0 | 0 | 0 | 0 | 0 |
| <ul> <li>d. I feel that this app is <u>appropriate</u> for military service members</li> </ul> | O | 0 | 0 | 0 | 0 |
| e. I would <u>recommend</u> this app to fellow <u>service members</u> | 0 | 0 | 0 | 0 | 0 |
| <ul> <li>I would <u>recommend</u> this app to a civilian<br/><u>friend</u></li> </ul> | 0 | 0 | 0 | 0 | 0 |
| g. This app helped me <u>understand</u> what prescription drug misuse is | 0 | 0 | 0 | 0 | 0 |
| The following questions are about specific sect | ions of the a | pp. | 2912121 | | |
| h. The My Meds section was useful | 0 | 0 | 0 | 0 | 0 |
| i. The Assessment section was useful | 0 | 0 | 0 | 0 | 0 |
| j. The Practice section was useful | 0 | 0 | 0 | 0 | 0 |
| k. The Learn section was useful | 0 | 0 | 0 | 0 | 0 |
| I. The Recommendations section was useful | 0 | 0 | 0 | 0 | 0 |
| m. The Resources section was useful | 0 | 0 | 0 | 0 | 0 |
| n. The Logbook section was useful | 0 | 0 | 0 | 0 | 0 |
| o. Other TBD section | 0 | 0 | 0 | 0 | 0 |
| p. Other TBD section | 0 | 0 | 0 | APPROVED | 9 |
| Vomine Date: 14 MAV 2019 | G-29 | | DATE: | 9 1 4 1 8<br>9 1 4 1 1 9<br>h Research Center 8 | In Diego |

| 35. | What did you like best about the app? |
|---|---|
| 36. | What did you like <u>least</u> about the app? |
| <b>37</b> . | What suggestions do you have for improving the app? |
| | How much technical difficulty did you experience with this app? O No technical difficulty O Very little technical difficulty O Some technical difficulty O Quite a bit technical difficulty O Nearly constant technical difficulty |
| 39. | Would you rather have gotten the information from this app in a different format? O Yes (What other format?) O No |
| | How much total time did you spend using this app over the past 1 month? I did not use the app 1-15 minutes 16-30 minutes 31-60 minutes Between 1 to 2 hours Between 2 to 3 hours Between 3 to 4 hours More than 4 hours |
| | How frequently did you use the app on average over the past 1 month? I did not use the app About once a month Several times a month Once a week Several times a week About once a day Several times a day |

#### **SUBMIT SURVEY**

Thanks for completing this survey! We greatly appreciate your participation!



## [Online]

# Prescription Drug Awareness Survey

1-month posttest (control group)

Protocol # NHRC.2016.0019

Naval Health Research Center

140 Sylvester Rd.

San Diego, CA 92106-3521

APPROVED

DATE: 6 1 4 1 16

EXP: 6 14 1 19

Naval Health Research Center San Diego

| OGIN |
|---------|
| f If-IN |

Please enter your non-DoD email address.

(Your email is the login for the surveys. This information will <u>not</u> be used for any other purpose. Once surveys are collected and linked together, your email address will be deleted from the study.)

Your E-mail address:


APPROVED

DATE: 6 1 41 /8 JU

EXP: 6 1/4 | 19

Naval Health Research Center San Diego

#### **MEDICATION AND PAIN**

## 1. Please answer the following.

| | | No | Yes |
|---|---|---|---|
| h. | Are you currently taking a prescription medication? | 0 | 0 |
| i. | Are you currently taking a prescription PAIN medication? | 0 | 0 |
| j. | Are you currently taking a prescription medication other than a pain medication? | 0 | 0 |
| k. | Are all of your prescriptions filled through the same pharmacy system? | 0 | 0 |
| l. | Have you experienced an illness or injury for which you are currently being treated? | 0 | 0 |
| m. | Have you experienced an illness or injury for which you still experience chronic pain? | 0 | 0 |
| n. | Are you currently experiencing pain? | 0 | 0 |

#### **TAKING MEDICATION IN GENERAL**

#### 2. Please indicate how often the following has happened to you...

| | | Never | Occasionally | Sometimes | Often | Always |
|---|---|---|---|---|---|---|
| g. | At times I need to borrow pain medication from friends or family to get relief | 0 | 0 | 0 | 0 | 0 |
| h. | I get pain medication from more<br>than one doctor in order to have<br>enough medication for my pain | 0 | 0 | 0 | 0 | 0 |
| i. | At times I need to take medication more often than it is prescribed in order to relieve my pain | 0 | 0 | 0 | 0 | 0 |
| j. | How many times in the <u>past year</u> have you asked your doctor to increase your prescribed dosage of pain medication in order to get relief? | 0 | 0 | 0 | 0 | 0 |
| k. | How many times in the <u>past year</u> have you run out of pain medication early and had to request an early refill? | 0 | 0 | 0 | 0 | 0 |
| l. | How many times in the <u>past year</u> have you accidentally misplaced your prescription for pain medication and had to ask for another? | 0 | 0 | 0 | 0 | 0 |

G-33


APPROVED

DATE: 6 1 4 1 /8 10

EXP: 6 1/4 1 /9

Naval Health Research Center San Diego

#### **MEDICATION LAST 30 DAYS**

3. Please answer each question as honestly as possible regarding the <u>past 30 days</u>. There are no right or wrong answers. If you are unsure about how to answer the question, please give the best answer you can.

| • | Never | Seldom | Sometimes | Often | Very<br>often |
|---|---|---|---|---|---|
| r. In the past 30 days, how often have you had trouble with thinking clearly or had memory problems? | 0 | 0 | 0 | 0 | 0 |
| s. In the past 30 days, how often do people<br>complain that you are not completing<br>necessary tasks? (i.e., doing things that<br>need to be done, such as going to class,<br>work or appointments) | 0 | 0 | 0 | 0 | 0 |
| t. In the past 30 days, how often have you had to go to someone other than your prescribing physician to get sufficient pain relief from medications? (i.e., another doctor, the Emergency Room, friends, street sources) | O | 0 | 0 | 0 | 0 |
| u. In the past 30 days, how often have you<br>taken your medications differently from<br>how they are prescribed? | 0 | 0 | 0 | 0 | 0 |
| v. In the past 30 days, how often have you seriously thought about hurting yourself? | 0 | 0 | 0 | 0 | 0 |
| w.In the past 30 days, how much of your<br>time was spent thinking about opioid<br>medications (having enough, taking<br>them, dosing schedule, etc.)? | 0 | 0 | 0 | 0 | 0 |
| x. In the past 30 days, how often have you been in an argument? | 0 | 0 | 0 | 0 | 0 |
| y. In the past 30 days, how often have you<br>had trouble controlling your anger (e.g.,<br>road rage, screaming, yelling, etc.)? | 0 | 0 | 0 | 0 | 0 |


APPROVED

DATE: 6 14 18

EXP: 6 1/4 19

Naval Health Research Center San Diego

| z. In the past 30 days, how often have you needed to take pain medications belonging to someone else? aa. In the past 30 days, how often have you been worried about how you're handling your medications? Never Seldom Sometimes Often Very often bb. In the past 30 days, how often have others been worried about how you're handling your medications? cc. In the past 30 days, how often have you had to make an emergency phone call or show up at the clinic without an appointment? dd. In the past 30 days, how often have you had to take more of your medication on than prescribed? ff. In the past 30 days, how often have you borrowed pain medicato from someone else? gg. In the past 30 days, how often have you used your pain medicine for symptoms other than for pain (e.g., to help you sleep, improve your mood, or relieve stress)? hh. In the past 30 days, how often have you had to visit the Emergency Room? | | | 8 Land | nar App, r rotocor | | 0.0012 |
|---|---|---|---|---|---|---|
| been worried about how you're handling your medications? Never Seldom Sometimes Often Very often bb. In the past 30 days, how often have others been worried about how you're handling your medications? cc. In the past 30 days, how often have you had to make an emergency phone call or show up at the clinic without an appointment? dd. In the past 30 days, how often have you gotten angry with people? ee. In the past 30 days, how often have you had to take more of your medication than prescribed? ff. In the past 30 days, how often have you borrowed pain medication from someone else? gg. In the past 30 days, how often have you used your pain medicine for symptoms other than for pain (e.g., to help you sleep, improve your mood, or relieve stress)? hh. In the past 30 days, how often have you O O O O O O O O O O O O O O O O O O | needed to take pain medications | 0 | 0 | 0 | 0 | 0 |
| bb. In the past 30 days, how often have others been worried about how you're handling your medications? cc. In the past 30 days, how often have you had to make an emergency phone call or show up at the clinic without an appointment? dd. In the past 30 days, how often have you gotten angry with people? ee. In the past 30 days, how often have you had to take more of your medication than prescribed? ff. In the past 30 days, how often have you borrowed pain medication from someone else? gg. In the past 30 days, how often have you used your pain medicine for symptoms other than for pain (e.g., to help you sleep, improve your mood, or relieve stress)? hh. In the past 30 days, how often have you | been worried about how you're | 0 | 0 | 0 | 0 | 0 |
| others been worried about how you're handling your medications? cc. In the past 30 days, how often have you had to make an emergency phone call or show up at the clinic without an appointment? dd. In the past 30 days, how often have you gotten angry with people? ee. In the past 30 days, how often have you had to take more of your medication than prescribed? ff. In the past 30 days, how often have you borrowed pain medication from someone else? gg. In the past 30 days, how often have you used your pain medicine for symptoms other than for pain (e.g., to help you sleep, improve your mood, or relieve stress)? hh. In the past 30 days, how often have you O O O O O O O O O O O O O O O O O O O | | Never | Seldom | Sometimes | Often | • |
| had to make an emergency phone call or show up at the clinic without an appointment? dd. In the past 30 days, how often have you gotten angry with people? ee. In the past 30 days, how often have you had to take more of your medication than prescribed? ff. In the past 30 days, how often have you borrowed pain medication from someone else? gg. In the past 30 days, how often have you used your pain medicine for symptoms other than for pain (e.g., to help you sleep, improve your mood, or relieve stress)? hh. In the past 30 days, how often have you | others been worried about how you're | 0 | 0 | 0 | 0 | 0 |
| gotten angry with people? ee. In the past 30 days, how often have you had to take more of your medication than prescribed? ff. In the past 30 days, how often have you borrowed pain medication from someone else? gg. In the past 30 days, how often have you used your pain medicine for symptoms other than for pain (e.g., to help you sleep, improve your mood, or relieve stress)? hh. In the past 30 days, how often have you | had to make an emergency phone call or show up at the clinic without an | 0 | 0 | 0 | 0 | |
| had to take more of your medication than prescribed? ff. In the past 30 days, how often have you borrowed pain medication from someone else? gg. In the past 30 days, how often have you used your pain medicine for symptoms other than for pain (e.g., to help you sleep, improve your mood, or relieve stress)? hh. In the past 30 days, how often have you O | | 0 | 0 | 0 | 0 | 0 |
| borrowed pain medication from OOOOOOOOOOOOOOOOOOOOOOOOOOOOOOOOOOOO | had to take more of your medication | 0 | 0 . | 0 | 0 | 0 |
| used your pain medicine for symptoms other than for pain (e.g., to help you osleep, improve your mood, or relieve stress)? hh. In the past 30 days, how often have you ooo | borrowed pain medication from | 0 | 0 | 0 | 0 | 0 |
| | used your pain medicine for symptoms other than for pain (e.g., to help you sleep, improve your mood, or relieve | 0 | 0 | 0 | 0 | 0 |
| | | 0 | 0 | 0 | 0 | 0 |

#### HOUSEHOLD

#### 4. Please answer the following.

| | | No | Yes |
|---|---|---|---|
| d. | Do you live with others? | 0 | 0 |
| e. | Some types of medication pose a greater risk of misuse. These include some pain medications, benzodiazepines muscle relaxants, sleeping medications, and some anxiety medications among others. Is someone in your household or living quarters taking these types of medications? | 0 | 0 |
| f. | Have you shared your prescription medication with others? | 0 | 0 |
| | G-35 | | DATE: 6 14 1/8 00 |


APPROVED

DATE: 6 14 1/8 19

EXP: 6 1/4 1/9

Naval Health Research Center Sen Diego
## Please continue onto next page.

| | COMMUNI | CATION | | | |
|---|---|---|---|---|---|
| 5. If you wanted to, how <u>prepared</u> do you feel to talk to? | Very<br>unprepared | Somewhat unprepared | Neutral | Somewhat prepared | Very<br>prepared |
| e. Someone in your chain of command if you were concerned about YOUR possible misuse of a prescribed medication? | 0 | 0 | 0 | 0 | 0 |
| f. Your <u>doctor</u> if you were concerned<br>about <u>YOUR</u> possible misuse of a<br>prescribed medication? | 0 | 0 | 0 | 0 | 0 |
| g. A <u>buddy</u> (fellow service member) if you were concerned about <u>THEIR</u> possible misuse of a prescribed medication? | 0 | 0 | 0 | 0 | 0 |
| h. A <u>spouse</u> (or significant other) if you were concerned about <u>THEIR</u> possible misuse of a prescribed medication? | 0 | O 2 | 0 | 0 | 0 |
| | ATTITU | DES | | | |

#### 9. Please indicate how much you agree or disagree with the statements.

| | | Strongly<br>disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Strongly<br>agree |
|---|---|---|---|---|---|---|
| w. | Misusing prescription drugs is dangerous. | 0 | 0 | 0 | 0 | 0 |
| х. | Most service members misuse prescription drugs at some point while on active duty. | 0 | 0 | 0 | 0 | 0 |
| y. | It's not a big deal to share prescription medication with someone if you're trying to help them. | 0 | 0 | 0 | 0 | 0 |
| z. | It should be illegal to share prescription medication with friends. | 0 | 0 | 0 | 0 | 0 |

G-36


APPROVED

DATE: 6 1 4 1 /8

EXP: 6 1 /4 1 /9

Naval Health Research Center San Diego

#### Hurtado, Evaluation of a Drug Abuse Educational App, Protocol # NHRC.2016.0019

| nunado, Evaluad | ion of a Diug A | touse Education | at App, Frotoco | # NIIKC.201 | 0.0019 |
|---|---|---|---|---|---|
| aa. It should be illegal to share prescription medication with family members. | 0 | 0 | 0 | 0 | 0 |
| bb. If you've been prescribed medication by<br>your doctor, you should take it only as<br>directed. | 0 | 0 | 0 | 0 | 0 |
| cc. If you share your prescription medications with friends or family, you are putting their health at risk. | 0 | 0 | 0 | 0 | 0 |
| | Strongly<br>disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Strongly<br>agree |
| dd. The risk of getting in trouble for taking pain medication differently than prescribed is a concern for me. | 0 | 0 | 0 | 0 | 0 |
| ee. There is a high risk of getting caught if you take your own old prescription medication. | 0 | 0 | 0 | 0 | 0 |
| ff. Using someone else's prescription medication can be hazardous to your health. | 0 | 0 | 0 | 0 | 0 |
| gg. Using someone else's prescription medication can cost you your military career. | 0 | 0 | 0 | 0 | 0 |
| hh. It is no big deal if I take a higher dose of<br>my prescription pain reliever than<br>directed. | 0 | 0 | 0 | 0 | 0 |
| ii. It is risky to my health to take my medication more often than prescribed. | 0 | 0 | 0 | 0 | 0 |
| jj. Even if a medication label says not to take<br>it with alcohol, it is ok to take it with only<br>one drink. | 0 | 0 | 0 | 0 | 0 |
| kk. Drinking alcohol with prescription pain relievers is only risky if you are binge drinking. | 0 | 0 | 0 | 0 | 0 |
| II. If I have questions about a prescription<br>medication, I should ask my provider. | 0 | 0 | 0 | 0 | 0 |
| mm. If I have questions about a prescription medication, I should ask the pharmacy tech. | 0 | 0 | 0 | 0 | 0 |
| nn. It is important to read the label on my prescription medication. | 0 | 0 | 0 | 0 | 0 |
| oo. It is important to read the material that the pharmacy provides with my prescription medication. | 0 | 0 | 0 | 0 | 0 |

G-37

APPROVED

DATE: 6 14 1/8 TD

EXP: 6 114 1 19

Naval Health Research Center San Diego

#### Hurtado, Evaluation of a Drug Abuse Educational App, Protocol # NHRC.2016.0019 pp. If I have concerns about my medication, 0 O 0 0 it's important that I know where to go for information. qq. It is ok to use your leftover prescription 0 0 0 0 0 medication for a new condition. rr. There is nothing wrong with taking an 0 0 0 0 0 extra dose of my prescription pain reliever if I am in pain.

### 10. Please indicate how much you agree or disagree with the statements.

| | | Strongly<br>disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Strongly<br>agree |
|---|---|---|---|---|---|---|
| i. | There are certain situations where it is ok to take someone else's prescribed medication. | 0 | 0 | 0 | 0 | 0 |
| j. | If a person is in physical pain from an injury, taking someone else's prescription medication is okay. | 0 | 0 | 0 | 0 | 0 |
| k. | As long as it makes you feel better and not worse, it's fine to take prescription drugs while drinking. | 0 | 0 | 0 | 0 | 0 |
| l. | An individual should only take medication that is prescribed to them by a medical professional. | 0 | 0 | 0 | 0 | 0 |
| m. | It is acceptable for a fellow service member to borrow someone's prescription medication in order to enhance their readiness. | 0 | 0 | 0 | 0 | 0 |
| n. | It is ok for a service member to take medication that is not prescribed to them in order to decrease appetite and lose weight. | 0 | 0 | 0 | 0 | 0 |
| 0. | Using prescribed medications to stay awake for duty is okay. | 0 | 0 | 0 | 0 | 0 |


DATE: 6 1411

Naval Health Research Center San Diego

| Hurtado, Evaluation of a Dr | ug Abuse Educ | ational App, Prot | ocol # NHRC.2 | 016.0019 |
|---|---|---|---|---|
| p. Taking medication that is not prescribed to you should be illegal. | 0 | 0 | 0 | 0 |
| 11. How much do you think people <u>risk harming the</u> | mselves (ph | ysically or in o | ther ways) b | y? |
| | No risk | Slight risk | Moderate<br>risk | Great risk |
| f. Taking <u>someone else's</u> prescription drug (examples: oxycodone, Valium)? | 0 | 0 | 0 | 0 |
| g. Taking a prescription drug (examples: oxycodone,<br>Valium) in <u>higher doses</u> than what a doctor<br>prescribed? | 0 | 0 | 0 | 0 |
| h. Taking a prescription drug (examples: oxycodone, Valium) together with alcohol or other drugs? | 0 | 0 | 0 | 0 |
| i. Having 5 or more drinks of alcohol once or twice each weekend? | 0 | 0 | 0 | 0 |
| j. Smoking marijuana regularly (more than once a week)? | 0 | 0 | 0 | 0 |
| 9. Please indicate how much you agree or disagree v | with the stat | ements. | | |
| | Strongly<br>disagree | Disagree | Agree | Strongly agree |
| e. I have made a final decision to stay away from<br>misusing prescription drugs (examples:<br>oxycodone, Valium). | 0 | 0 | 0 | 0 |
| f. I have made a final decision to stay away from abusing prescription drugs (examples: oxycodone, Valium). | 0 | 0 | 0 | 0 |
| g. I intend to use my prescription medications exactly as prescribed by my provider. | 0 | 0 | 0 | 0 |
| h. I plan to intervene if I see someone misusing prescription medication. | 0 | 0 | 0 | 0 |


APPROVED

DATE: 6 14 118 J.D

EXP: 6 114 1 19

Navai Health Research Center San Diego

#### KNOWLEDGE

- 33. Based upon DoD policy, which of the following is NOT an example of prescription drug misuse?
- f. Taking more of your medication that is prescribed
- g. Taking your medication at 2150 instead of 2200 because you plan to go to sleep
- h. Using the prescription you got earlier this year for your knee for a back strain you got this week
- i. Taking your pain medication 4 times a day instead of 3 like it says on the label
- j. Giving some of your medication to your spouse because he or she ran out
- **34.** Which of the following is <u>NOT</u> a recommendation in the Prescription for Discharge campaign to protect Sailors and Marines from prescription drug misuse/abuse?
- f. Report promptly
- g. Take correctly
- h.Save for emergencies
- i. Never share
- j. Dispose properly
- **35.** What should a service member do if they receive a prescription medication from a *non-military* medical treatment facility?
- f. Report it to the Chaplain
- g. It ONLY needs to be reported to their military health care provider if they had an adverse reaction
- h.It does not need to be reported
- i. Report it to their military health care provider at their next visit
- j. Report it to their chain of command and ensure it is entered into their military health record
- 36. What type of alternative treatment involves visualizing specific positive scenes to reduce stress?
- f. Biofeedback
- g. Acupuncture
- h.Yoga
- i. Guided Imagery
- j. Physical Therapy
- 37. What type of alternative treatment involves becoming mindful of one's thoughts and sensations in a nonjudgmental way?
- f. Physical Therapy
- g. Biofeedback
- h.Chiropractic Therapies
- i. Massage Therapy
- j. Meditation
- **38.** What can you do if you suspect someone is misusing prescription medication?
- f. Provide support
- g. Be a role model
- h. Keep medications safe and secured


- i. Inform chain of command or law enforcement officials
- j. All of the above
- **39.** Which of the following is <u>NOT</u> potentially a sign or symptom associated with prescription drug misuse?

APPROVED

DATE: 6 14 1 18

EXP: 6 14 1 19

Naval Health Research Center San Diego

- f. Relationship problems
- g. Sudden weight loss or gain
- h. Asking your doctor questions about your prescription
- i. Changes in appetite or sleep patterns
- j. Decreased performance at work
- 40. What are the two most commonly misused prescription drugs among military personnel?
  - e. Pain relievers (opioids) and central nervous system depressants (sedatives)
  - f. Pain relievers (opioids) and protease inhibitors
  - g. Central nervous system depressants (sedatives) and protease inhibitors
  - h.Central nervous system depressants (sedatives) and central nervous system stimulants Pain relievers (opioids) and central nervous system stimulants
- 41. Which of the following is a negative consequence of misusing prescription drugs?
  - f. Drug addiction
  - g. Altered judgment
  - h.Unintentional overdose
  - i. Drug tolerance
  - j. All of the above
- **42.** What is a specific sign or symptom of prescription drug misuse?
  - f. Faking illness or injury to obtain medications
  - g. Excessive visits to the doctor
  - h. Stealing, forging, or selling prescriptions
  - i. None of the above
  - j. All of the above

DATE: 6 14 1/8 DEXP: 6 1/4/1/9

- **43.** Which of the following could help you reduce your risk of prescription drug misuse? (Select the best answer)
  - f. Ask your friend which medication worked best for them to treat pain
  - g. Take your old prescription for pain without consulting your doctor
  - h. Wait until your pain is unbearable before taking pain medication instead of taking it at the regular intervals indicated
  - i. Talk to your doctor about symptoms you may be having or concerns about your medication
  - j. Mix your prescription medication with over-the-counter medicine and supplements
- 44. It is important to talk to your doctor or pharmacist about... (Select the best answer)
  - f. Using over-the-counter medications while using your prescription
  - g. Supplements that you routinely take
  - h. Symptoms and side effects you are experiencing
  - i. A and C
  - i. All of the above
- 45. TRUE OR FALSE: Everyday activities such as playing sports cannot cause traumatic brain injuries (TBI).
  - c. TRUE
  - d.FALSE
- **46.** TRUE OR FALSE: Prescription drugs are regulated so they are always safe to take.
  - c. TRUE
  - d.FALSE
- **47.** TRUE OR FALSE: It is safe to take prescription medication from a previous health problem to treat new symptoms.
  - c. TRUE
  - d.FALSE
- **48.** Which of the following is a good resource for someone seeking information about a prescription medication misuse problem? (Select all that apply)
- f. SACO or DAPA
- g. Corpsman or other medical provider
- h.Commanding Officer
- i. Diversity Officer
- j. MilitaryOneSource
- 49. Drinking alcohol with prescription medication can do which of the following? (Select all that apply)
  - f. Increase side effects
  - g. Increase effectiveness
  - h.Decrease effectiveness
  - i. Decrease sedative effects
  - j. Increase risk of a toxic reaction


DATE: 6/4/8
EXP: 6/4/9
Naval Health Research Center San Diego

- **50.** Which of the following has contributed to the increase in prescription drug abuse among service members? (Select all that apply)
  - f. Increase in prescriptions for pain related to injuries among OIF and OEF veterans
  - g. Decrease in military pharmacy regulations
  - h.Increase in average working hours among service members
  - i. Decrease in the number of compounds tested in drug screening
  - j. Increase in the number of military health care providers
- 51. Which step(s) can you take to reduce prescription drug misuse? (Select all that apply)
  - f. Use previously prescribed medication for a current health issue
  - g. Keep your medications safe and secured
  - h.Only borrow prescription medication from a spouse or other trusted source
  - i. Dispose of unused or expired prescription medication properly
  - j. Do not share medication
- **52.** Which of the following are key points you would want to discuss with your pharmacist when getting a new prescription? (Select all that apply)
  - f. Best time of day to take medication
  - g. Other health conditions the medication may be used for in the future
  - h.Prescribed dosage
  - i. Potential side effects and warnings
  - j. Alternative non-medical treatments
- 53. Which of the following are signs and symptoms of depression? (Select all that apply)
  - f. Changes in appetite or weight
  - g. Increased motivation
  - h.Increased energy
  - i. Decreased energy
  - j. Irritability
- 54. Which of the following statement(s) about sleep is TRUE? (Select all that apply)
  - f. The quality of sleep you are getting is just as important as the amount
  - g. Sleep problems can be a side effect of some medications
  - h. The amount of sleep you are getting is the most important aspect of sleep
  - i. Sleep problems can be a symptom of a mental health condition
  - j. Catching-up on sleep is just as effective as regular sleep
- **55.**What are two common forms of treatment for mental health conditions such as depression, anxiety, and PTSD? (Select all that apply)
  - f. Medication
  - g. Physical therapy
  - h. Dietary changes
  - i. No treatment available


j. Psychotherapy

**SUBMIT SURVEY** 

Thanks for completing this survey! We greatly appreciate your participation

EXP: 6 1/4 1 /9

# [Online]

# Prescription Drug Awareness Survey

3-month posttest (intervention group)

Protocol # NHRC.2016.0019
Naval Health Research Center
140 Sylvester Rd.
San Diego, CA 92106-3521

APPROVED

DATE: 6 14 18

EXP: 6 14 19

Naval Health Research Center San Diego

#### LOGIN

Please enter your non-DoD email address.

(Your email is the login for the surveys. This information will <u>not</u> be used for any other purpose. Once surveys are collected and linked together, your email address will be deleted from the study.)

Your E-mail address:

| 170 |
|-----|

APPROVED

DATE: 6 141/8

EXP: 6 141/9

Naval Health Research Center San Diego

#### **MEDICATION AND PAIN**

#### 1. Please answer the following.

| | | No | Yes |
|---|---|---|---|
| 0. | Are you currently taking a prescription medication? | 0 | 0 |
| p. | Are you currently taking a prescription PAIN medication? | 0 | 0 |
| q. | Are you currently taking a prescription medication other than a pain medication? | 0 | 0 |
| r. | Are all of your prescriptions filled through the same pharmacy system? | 0 | 0 |
| s. | Have you experienced an illness or injury for which you are currently being treated? | 0 | 0 |
| t. | Have you experienced an illness or injury for which you still experience chronic pain? | 0 | 0 |
| u. | Are you currently experiencing pain? | 0 | 0 |

#### **TAKING MEDICATION IN GENERAL**

#### 2. Please indicate how often the following has happened to you...

| | | Never | Occasionally | Sometimes | Often | Always |
|---|---|---|---|---|---|---|
| m. | At times I need to borrow pain medication from friends or family to get relief | 0 | 0 | 0 | 0 | 0 |
| n. | I get pain medication from more than one doctor in order to have enough medication for my pain | 0 | 0 | 0 | 0 | 0 |
| 0. | At times I need to take medication more often than it is prescribed in order to relieve my pain | 0 | 0 | 0 | 0 | 0 |
| p. | How many times in the <u>past year</u> have you asked your doctor to increase your prescribed dosage of pain medication in order to get relief? | 0 | 0 | 0 | 0 | 0 |
| q. | How many times in the <u>past year</u> have you run out of pain medication early and had to request an early refill? | 0 | 0 | 0 | 0 | 0 |
| r. | How many times in the <u>past year</u> have you accidentally misplaced your prescription for pain medication and had to ask for another? | 0 | 0 | 0 | 0 | 0 |

APPROVED

DATE: 6 1 4 1 / 8 10

EXP: 6 1 / 4 / 9

Naval Health Research Center San Diego

## **MEDICATION LAST 30 DAYS**

3. Please answer each question as honestly as possible regarding the past 30 days. There are no right or wrong answers. If you are unsure about how to answer the question, please give the best answer you can.

| | Never | Seldom | Sometimes | Often | Very<br>often |
|---|---|---|---|---|---|
| ii. In the past 30 days, how often have you had trouble with thinking clearly or had memory problems? | 0 | 0 | 0 | 0 | 0 |
| jj. In the past 30 days, how often do people<br>complain that you are not completing<br>necessary tasks? (i.e., doing things that<br>need to be done, such as going to class,<br>work or appointments) | 0 | 0 | 0 | 0 | 0 |
| kk. In the past 30 days, how often have you had to go to someone other than your prescribing physician to get sufficient pain relief from medications? (i.e., another doctor, the Emergency Room, friends, street sources) | 0 | 0 | 0 | 0 | 0 |
| II. In the past 30 days, how often have you<br>taken your medications differently from<br>how they are prescribed? | 0 | 0 | 0 | 0 | 0 |
| mm. In the past 30 days, how often have you seriously thought about hurting yourself? | 0 | 0. | 0 | 0 | 0 |
| nn. In the past 30 days, how much of<br>your time was spent thinking about<br>opioid medications (having enough,<br>taking them, dosing schedule, etc.)? | 0 | 0 | 0 | 0 | 0 |
| oo. In the past 30 days, how often have you been in an argument? | 0 | 0 | 0 | 0 | 0 |
| pp. In the past 30 days, how often have you<br>had trouble controlling your anger (e.g.,<br>road rage, screaming, yelling, etc.)? | 0 | 0 | 0 | 0 | 0 |
| qq. In the past 30 days, how often have you needed to take pain medications belonging to someone else? | 0 | 0 | 0 | 0 | 0 |
| rr. In the past 30 days, how often have you been worried about how you're handling your medications? Version Date14 MAY 2018 | O<br>G-47 | 0 | DATE: <u>6</u> /<br>EXP: <u>6</u> / | PROVED 41/8 141/9 earch Center San | Jr.D<br>Diego |

#### Hurtado, Evaluation of a Drug Abuse Educational App, Protocol # NHRC.2016.0019

| | Never | Seldom | Sometimes | Often | Very<br>often |
|---|---|---|---|---|---|
| ss. In the past 30 days, how often have others been worried about how you're handling your medications? | 0 | 0 | 0 | 0 | 0 |
| tt. In the past 30 days, how often have you had to make an emergency phone call or show up at the clinic without an appointment? | 0 | 0 | 0 | 0 | 0 |
| uu. In the past 30 days, how often have you gotten angry with people? | 0 | 0 | 0 | 0 | 0 |
| vv. In the past 30 days, how often have you<br>had to take more of your medication<br>than prescribed? | 0 | 0 | 0 | 0 | 0 |
| ww. In the past 30 days, how often have you borrowed pain medication from someone else? | 0 | 0 | 0 | 0 | 0 |
| xx. In the past 30 days, how often have you used your pain medicine for symptoms other than for pain (e.g., to help you sleep, improve your mood, or relieve stress)? | 0 | 0 | 0 | 0 | 0 |
| yy. In the past 30 days, how often have you had to visit the Emergency Room? | 0 | 0 | 0 | 0 | 0 |

#### HOUSEHOLD

#### 4. Please answer the following.

| | | No | Yes |
|---|---|---|---|
| g. | Do you live with others? | 0 | 0 |
| h. | Some types of medication pose a greater risk of misuse. These include some pain medications, benzodiazepines muscle relaxants, sleeping medications, and some anxiety medications among others. Is someone in your household or living quarters taking these types of medications? | 0 | 0 |
| i. | Have you shared your prescription medication with others? | 0 | 0 |

Please continue onto next page.

APPROVED

DATE: 6 14 1 /8

EXP: 6 1/4/19

Naval Health Research Center San Diego

#### COMMUNICATION Very Somewhat 5. If you wanted to, how prepared do Somewhat Very unprepared unprepared Neutral prepared prepared you feel to talk to ...? i. Someone in your chain of command 0 0 0 0 0 if you were concerned about YOUR possible misuse of a prescribed medication? j. Your doctor if you were concerned 0 0 0 0 0 about YOUR possible misuse of a prescribed medication? k. A buddy (fellow service member) if 0 0 0 0 0 you were concerned about THEIR possible misuse of a prescribed medication? I. A spouse (or significant other) if you 0 0 0 0 0 were concerned about THEIR possible misuse of a prescribed medication? **ATTITUDES**

#### 12. Please indicate how much you agree or disagree with the statements.

| | Strongly<br>disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Strongly<br>agree |
|---|---|---|---|---|---|
| ss. Misusing prescription drugs is dangerous. | 0 | 0 | 0 | 0 | 0 |
| tt. Most service members misuse prescription drugs at some point while on active duty. | 0 | 0 | 0 | 0 | 0 |
| uu. It's not a big deal to share prescription medication with someone if you're trying to help them. | 0 | 0 | 0 | 0 | 0 |
| vv. It should be illegal to share prescription medication with friends. | 0 | 0 | 0 | 0 | 0 |
| ww. It should be illegal to share prescription medication with family members. | 0 | 0 | 0 | 0 | 0 |
| your doctor, you should take it only as directed. | 0 | 0 | 0 | 0 | 0 |
| yy. If you share your prescription medications with friends or family, you are putting their health at risk. | 0 | 0 | 0 | 0 | 0 |
| | | 11 | | PPROVED 18 | 70 |

G-49

#### Hurtado, Evaluation of a Drug Abuse Educational App, Protocol # NHRC.2016.0019

| riuriado, Evalua | | | ai App, Protocoi | | |
|---|---|---|---|---|---|
| | Strongly<br>disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Strongly<br>agree |
| zz. The risk of getting in trouble for taking<br>pain medication differently than<br>prescribed is a concern for me. | 0 | 0 | 0 | 0 | 0 |
| aaa. There is a high risk of getting caught if you take your own old prescription medication. | 0 | 0 | 0 | 0 | 0 |
| bbb. Using someone else's prescription<br>medication can be hazardous to your<br>health. | 0 | 0 | 0 | 0 | 0 |
| ccc. Using someone else's prescription medication can cost you your military career. | 0 | 0 | 0 | 0 | 0 |
| ddd. It is no big deal if I take a higher dose<br>of my prescription pain reliever than<br>directed. | 0 | 0 | 0 | 0 | 0 |
| eee. It is risky to my health to take my medication more often than prescribed. | 0 | 0 | 0 | 0 | 0 |
| fff. Even if a medication label says not to take it with alcohol, it is ok to take it with only one drink. | 0 | 0 | 0 | 0 | 0 |
| ggg. Drinking alcohol with prescription pain relievers is only risky if you are binge drinking. | 0 | 0 | 0 | 0 | 0 |
| hhh. If I have questions about a prescription medication, I should ask my provider. | 0 | 0 | 0 | 0 | 0 |
| iii. If I have questions about a prescription medication, I should ask the pharmacy tech. | 0 | 0 | 0 | 0 | 0 |
| jjj. It is important to read the label on my prescription medication. | 0 | 0 | 0 | 0 | 0 |
| kkk. It is important to read the material that the pharmacy provides with my prescription medication. | 0 | 0 | 0 | 0 | 0 |
| III. If I have concerns about my medication,<br>it's important that I know where to go for<br>information. | 0 | 0 | 0 | 0 | 0 |
| mmm. It is ok to use your leftover prescription medication for a new condition. | 0 | 0 | 0 | 0 | 0 |
| nnn. There is nothing wrong with taking an extra dose of my prescription pain reliever if I am in pain. | 0 | 0 | 0 | 0 | 0 |

APPROVED

DATE: 6 1418

EXP: 6 1419

Naval Health Research Center San Diego

### 13. Please indicate how much you agree or disagree with the statements.

| | | Strongly<br>disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Strongly<br>agree |
|---|---|---|---|---|---|---|
| q. | There are certain situations where it is ok to take someone else's prescribed medication. | 0 | 0 | 0 | 0 | 0 |
| r. | If a person is in physical pain from an injury, taking someone else's prescription medication is okay. | 0 | . 0 | 0 | 0 | 0 |
| S. | As long as it makes you feel better and not worse, it's fine to take prescription drugs while drinking. | 0 | 0 | 0 | 0 | 0 |
| t. | An individual should only take medication that is prescribed to them by a medical professional. | 0 | 0 | 0 | 0 | 0 |
| u. | It is acceptable for a fellow service member to borrow someone's prescription medication in order to enhance their readiness. | 0 | 0 | 0 | 0 | 0 |
| v. | It is ok for a service member to take medication that is not prescribed to them in order to decrease appetite and lose weight. | 0 | 0 | 0 | 0 | 0 |
| w. | Using prescribed medications to stay awake for duty is okay. | 0 | 0 | 0 | 0 | 0 |
| x. | Taking medication that is not prescribed to you should be illegal. | 0 | 0 | 0 | 0 | 0 |

# 14. How much do you think people <u>risk harming themselves</u> (physically or in other ways) by...?

| | No risk | Slight risk | Moderate<br>risk | Great risk |
|---|---|---|---|---|
| k. Taking <u>someone else's</u> prescription drug (examples: oxycodone, Valium)? | 0 | 0 | 0 | 0 |
| | 2 | DATE: | PPROVED | nD |
| G-51 rsion Date14 MAY 2018 | | EXP: 6 | 114 1 19<br>Research Center Sar | n Diego |

| Hurtado, Evaluation of a Di | rug Abuse Educ | ational App, Pro | tocol # NHRC | 2.2016.0019 |
|---|---|---|---|---|
| I. Taking a prescription drug (examples: oxycodone,<br>Valium) in <u>higher doses</u> than what a doctor<br>prescribed? | 0 | 0 | 0 | 0 |
| m.Taking a prescription drug (examples: oxycodone, Valium) together with alcohol or other drugs? | 0 | 0 | 0 | 0 |
| n. Having 5 or more drinks of alcohol once or twice each weekend? | 0 | 0 | 0 | 0 |
| o. Smoking marijuana regularly (more than once a week)? | 0 | 0 | 0 | 0 |
| 9. Please indicate how much you agree or disagree | with the stat | tements. | | |
| | Strongly disagree | Disagree | Agree | Strongly agree |
| i. I have made a final decision to stay away from<br>misusing prescription drugs (examples:<br>oxycodone, Valium). | 0 | 0 | 0 | 0 |
| <ul> <li>j. I have made a final decision to stay away from<br/>abusing prescription drugs (examples: oxycodone,<br/>Valium).</li> </ul> | 0 | 0 | 0 | 0 |
| k. I intend to use my prescription medications exactly as prescribed by my provider. | 0 | 0 | 0 | 0 |
| I. I plan to intervene if I see someone misusing prescription medication. | 0 | 0 | 0 | 0 |
| KNOWLE | DGE | | | |
| <ol> <li>Based upon DoD policy, which of the following is k. Taking more of your medication that is prescribed l. Taking your medication at 2150 instead of 2200 becaus m. Using the prescription you got earlier this year for yo n. Taking your pain medication 4 times a day instead of 3 o. Giving some of your medication to your spouse becaus</li> <li>Which of the following is NOT a recommendation in protect Sailors and Marines from prescription drug m k. Report promptly</li> </ol> | se you plan to<br>ur knee for a<br>like it says on<br>e he or she ra<br>the Prescript | go to sleep<br>back strain you<br>the label<br>n out<br>ion for Discharg | got this wee | ·k |

G-52

n. Never share

- o. Dispose properly
- **12.** What should a service member do if they receive a prescription medication from a *non-military* medical treatment facility?
- k. Report it to the Chaplain
- I. It ONLY needs to be reported to their military health care provider if they had an adverse reaction
- m. It does not need to be reported
- n.Report it to their military health care provider at their next visit
- o. Report it to their chain of command and ensure it is entered into their military health record
- 13. What type of alternative treatment involves visualizing specific positive scenes to reduce stress?
- k. Biofeedback
- I. Acupuncture
- m. Yoga
- n.Guided Imagery
- o. Physical Therapy
- 14. What type of alternative treatment involves becoming mindful of one's thoughts and sensations in a nonjudgmental way?
- k. Physical Therapy
- I. Biofeedback
- m. Chiropractic Therapies
- n. Massage Therapy
- o.Meditation
- 15. What can you do if you suspect someone is misusing prescription medication?
- k. Provide support
- I. Be a role model
- m. Keep medications safe and secured
- n.Inform chain of command or law enforcement officials
- o.All of the above
- 16. Which of the following is <u>NOT</u> potentially a sign or symptom associated with prescription drug misuse?
  - k. Relationship problems
  - Sudden weight loss or gain
  - m. Asking your doctor questions about your prescription
  - n. Changes in appetite or sleep patterns
  - o. Decreased performance at work
- 17. What are the two most commonly misused prescription drugs among military personnel?
  - i. Pain relievers (opioids) and central nervous system depressants (sedatives)
  - j. Pain relievers (opioids) and protease inhibitors
  - k. Central nervous system depressants (sedatives) and protease inhibitors
  - I. Central nervous system depressants (sedatives) and central nervous system stimulants
    Pain relievers (opioids) and central nervous system stimulants
- 18. Which of the following is a negative consequence of misusing prescription drugs?
  - k. Drug addiction
  - I. Altered judgment

APPROVED

DATE: 6 141/8 PD

EXP: 6 1/41/9

Naval Health Research Center San Diego

G-53

#### Hurtado, Evaluation of a Drug Abuse Educational App, Protocol # NHRC.2016.0019

- m. Unintentional overdose
- n.Drug tolerance
- o.All of the above
- **19.** What is a specific sign or symptom of prescription drug misuse?
  - k. Faking illness or injury to obtain medications
  - I. Excessive visits to the doctor
  - m. Stealing, forging, or selling prescriptions
  - n. None of the above
  - o.All of the above

APPROVED

DATE: 6 14 1 18

EXP: 6 1/4 1 19

Naval Health Research Center San Diego

- 20. Which of the following could help you reduce your risk of prescription drug misuse? (Select the best answer)
  - k. Ask your friend which medication worked best for them to treat pain
  - I. Take your old prescription for pain without consulting your doctor
  - m. Wait until your pain is unbearable before taking pain medication instead of taking it at the regular intervals indicated
  - n. Talk to your doctor about symptoms you may be having or concerns about your medication
  - o.Mix your prescription medication with over-the-counter medicine and supplements
- 21. It is important to talk to your doctor or pharmacist about... (Select the best answer)
  - k. Using over-the-counter medications while using your prescription
  - I. Supplements that you routinely take
  - m. Symptoms and side effects you are experiencing
  - n.A and C
  - o.All of the above
- 22. TRUE OR FALSE: Everyday activities such as playing sports cannot cause traumatic brain injuries (TBI).
  - e.TRUE
  - f. FALSE
- 23. TRUE OR FALSE: Prescription drugs are regulated so they are always safe to take.
  - e.TRUE
  - f. FALSE
- 24. TRUE OR FALSE: It is safe to take prescription medication from a previous health problem to treat new symptoms.
  - e.TRUE
  - f. FALSE
- 25. Which of the following is a good resource for someone seeking information about a prescription medication misuse problem? (Select all that apply)
- k. SACO or DAPA
- I. Corpsman or other medical provider
- m. Commanding Officer
- n.Diversity Officer
- o.MilitaryOneSource
- 26. Drinking alcohol with prescription medication can do which of the following? (Select all that apply)
  - k. Increase side effects
  - I. Increase effectiveness
  - m. Decrease effectiveness
  - n.Decrease sedative effects
  - o.Increase risk of a toxic reaction

APPROVED

DATE: 6 1 4 1 / 8

EXP: 6 1 14 1 / 9

Naval Health Research Cerrier San Diego

- 27. Which of the following has contributed to the increase in prescription drug abuse among service members? (Select all that apply)
  - k. Increase in prescriptions for pain related to injuries among OIF and OEF veterans
  - I. Decrease in military pharmacy regulations
  - m. Increase in average working hours among service members
  - n. Decrease in the number of compounds tested in drug screening
  - o.Increase in the number of military health care providers
- 28. Which step(s) can you take to reduce prescription drug misuse? (Select all that apply)
  - k. Use previously prescribed medication for a current health issue
  - I. Keep your medications safe and secured
  - m. Only borrow prescription medication from a spouse or other trusted source
  - n. Dispose of unused or expired prescription medication properly
  - o.Do not share medication
- 29. Which of the following are key points you would want to discuss with your pharmacist when getting a new prescription? (Select all that apply)
  - k. Best time of day to take medication
  - I. Other health conditions the medication may be used for in the future
  - m. Prescribed dosage
  - n. Potential side effects and warnings
  - o.Alternative non-medical treatments
- **30.** Which of the following are signs and symptoms of depression? (Select all that apply)
  - k. Changes in appetite or weight
  - I. Increased motivation
  - m. Increased energy
  - n. Decreased energy
  - o.Irritability
- **31.** Which of the following statement(s) about sleep is TRUE? (Select all that apply)
  - k. The quality of sleep you are getting is just as important as the amount
  - I. Sleep problems can be a side effect of some medications
  - m. The amount of sleep you are getting is the most important aspect of sleep
  - n. Sleep problems can be a symptom of a mental health condition
  - o. Catching-up on sleep is just as effective as regular sleep
- **32.** What are two common forms of treatment for mental health conditions such as depression, anxiety, and PTSD? (Select all that apply)
  - k. Medication
  - I. Physical therapy
  - m. Dietary changes
  - n.No treatment available
  - o.Psychotherapy



#### **RATINGS OF THE APP**

#### 33. Please rate the various aspects of the app.

| | | Disliked<br>very much | Disliked | Neither<br>liked nor<br>disliked | Liked | Liked very<br>much |
|---|---|---|---|---|---|---|
| d. | The app as a whole | 0 | 0 | 0 | 0 | 0 |
| e. | Overall content | 0 | 0 | 0 | 0 | 0 |
| f. | Overall appearance and graphics | 0 | 0 | 0 | 0 | 0 |

| 34. Please indicate how much you agree or d | isagree with | the stateme | ents. | | |
|---|---|---|---|---|---|
| | Strongly<br>disagree | Disagree | Neither agree nor disagree | Agree | Strongly<br>agree |
| a. The app was <u>useful</u> | 0 | 0 | 0 | 0 | 0 |
| q. I learned <u>new</u> information from this app | 0_ | 0 | 0 | 0 | 0 |
| r. The app was <u>easy</u> to use | 0 | 0 | 0 | 0 | 0 |
| <ul> <li>I feel that this app is appropriate for military service members</li> </ul> | 0 | 0 | 0 | 0 | 0 |
| t. I would <u>recommend</u> this app to fellow<br><u>service members</u> | 0 | 0 | 0 | 0 | 0 |
| <ul> <li>I would <u>recommend</u> this app to a civilian<br/><u>friend</u></li> </ul> | 0 | 0 | 0 | 0 | 0 |
| v. This app helped me <u>understand</u> what prescription drug misuse is | 0 | 0 | 0 | 0 | 0 |
| The following questions are about specific sect | ions of the a | pp. | | | |
| w. The My Meds section was useful | 0 | 0 | 0 | 0 | 0 |
| x. The Assessment section was useful | 0 | 0 | 0 | 0 | 0 |
| y. The Practice section was useful | 0 | 0 | 0 | 0 | 0 |
| z. The Learn section was useful | 0 | 0 | 0 | 0 | 0 |
| aa. The Recommendations section was useful | 0 | 0 | 0 | 0 | 0 |
| bb. The Resources section was useful | 0 | 0 | 0 | 0 | 0 |
| cc. The Logbook section was useful | 0 | 0 | 0 | 0 | 0 |
| dd. Other TBD section | O<br>G-57 | 0 | DATE: 6 / | ROVED 118 119 | |
| ersion Date14 MAY 2018 | | | Naval Health Res | earch Center San Dieg | 90 |

#### Hurtado, Evaluation of a Drug Abuse Educational App, Protocol # NHRC.2016.0019

Strongly agree

0

| | | Strongly<br>disagree | Disagree | Neither<br>agree nor<br>disagree | Agree |
|---|---|---|---|---|---|
| ee. O | Other TBD section | 0 | 0 | 0 | 0 |
| 36. W | /hat did you like <u>best</u> about the app?<br>/hat did you like <u>least</u> about the app? | | | | |
| 38. H<br>O<br>O<br>O | hat suggestions do you have for improvidow much technical difficulty did you expe<br>No technical difficulty<br>Very little technical difficulty<br>Some technical difficulty<br>Quite a bit technical difficulty<br>Nearly constant technical difficulty | | | | |
| 0 | ould you rather have gotten the informa Yes (What other format? No | | | erent format | ? |
| 00000000 | ow much total time did you spend using to I did not use the app 1-15 minutes 16-30 minutes 31-60 minutes Between 1 to 2 hours Between 2 to 3 hours Between 4 to 5 hours Between 4 to 5 hours Between 5-6 hours More than 6 hours | his app over | the <u>past 3 m</u> | onths? | |
| 000000 | ow frequently did you use the app on average I did not use the app One or two times during the past 3 more About once a month Several times a month Once a week Several times a week About once a day Several times a day | | past 3 mont | <u>hs</u> ? | |

DATE: 6 14 1 18

EXP: 6 14 1 19

Naval Health Research Center San Diego

#### **SUBMIT SURVEY**

Thanks for completing this survey! We greatly appreciate your participation!

APPROVED

DATE: 6 1 4 1 18

EXP: 6 114 1 19

Naval Health Research Center San Diego

# [Online]

# Prescription Drug Awareness Survey

3-month posttest (control group)

Protocol # NHRC.2016.0019

Naval Health Research Center

140 Sylvester Rd.

San Diego, CA 92106-3521

APPROVED

DATE: 6 14 1 18

EXP: 6 1 14 1 19

Navai Health Research Center San Diego

| | | | | | | | | | | LC | GIN | V | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Plea | se er | iter ' | your | non | -Do[ | ) em | ail a | ddre | ess. | | | | |
| | ır em<br>e sur<br>v.) | | | | | | | | | | | | • |
| 3100 | | •• | | | | | | | | | | | |
| You | r E-m | ail a | aare | <b>55.</b> | | | | | | | | | |
| You | r E-m | ail a | aare | 55. | | | ! | | | | | | Τ |

APPROVED

DATE: 6 14 1 18

EXP: 6 1/4 1 19

Naval Health Research Center San Diego

#### **MEDICATION AND PAIN**

### 1. Please answer the following.

| | No | Yes |
|---|---|---|
| v. Are you currently taking a prescription medication? | 0 | 0 |
| w. Are you currently taking a prescription PAIN medication? | 0 | 0 |
| x. Are you currently taking a prescription medication other than a pain medication? | 0 | 0 |
| y. Are all of your prescriptions filled through the same pharmacy<br>system? | 0 | 0 |
| z. Have you experienced an illness or injury for which you are currently being treated? | 0 | 0 |
| aa. Have you experienced an illness or injury for which you still<br>experience chronic pain? | 0 | 0 |
| bb. Are you currently experiencing pain? | 0 | 0 |

#### **TAKING MEDICATION IN GENERAL**

### 2. Please indicate how often the following has happened to you...

| | | Never | Occasionally | Sometimes | Often | Always |
|---|---|---|---|---|---|---|
| S. | At times I need to borrow pain medication from friends or family to get relief | 0 | 0 | 0 | 0 | 0 |
| t. | I get pain medication from more<br>than one doctor in order to have<br>enough medication for my pain | 0 | 0 | 0 | 0 | 0 |
| u. | At times I need to take medication more often than it is prescribed in order to relieve my pain | 0 | 0 | 0 | 0 | 0 |
| V. | How many times in the <u>past year</u> have you asked your doctor to increase your prescribed dosage of pain medication in order to get relief? | 0 | 0 | 0 | 0 | 0 |
| w. | How many times in the <u>past year</u> have you run out of pain medication early and had to request an early refill? | 0 | 0 | 0 | 0 | 0 |
| x. | How many times in the <u>past year</u> have you accidentally misplaced your prescription for pain medication and had to ask for another? | 0 | 0 | 0 | 0 | 0 |

DATE: 6 14 1 18

EXP: 6 1/4 1 19

Naval Health Research Center San Diego

G-62

#### **MEDICATION LAST 30 DAYS**

3. Please answer each question as honestly as possible regarding the <u>past 30 days</u>. There are no right or wrong answers. If you are unsure about how to answer the question, please give the best answer you can.

| | Never | Seldom | Sometimes | Often | Very<br>often |
|---|---|---|---|---|---|
| zz. In the past 30 days, how often have you had trouble with thinking clearly or had memory problems? | 0 | 0 | 0 | 0 | 0 |
| aaa. In the past 30 days, how often do people complain that you are not completing necessary tasks? (i.e., doing things that need to be done, such as going to class, work or appointments) | 0 | 0 | 0 | 0 | |
| bbb. In the past 30 days, how often have you had to go to someone other than your prescribing physician to get sufficient pain relief from medications? (i.e., another doctor, the Emergency Room, friends, street sources) | 0 | 0 | 0 | 0 | 0 |
| ccc. In the past 30 days, how often have<br>you taken your medications differently<br>from how they are prescribed? | 0 | 0 | 0 | 0 | 0 |
| ddd. In the past 30 days, how often have you seriously thought about hurting yourself? | 0 | 0 | 0 | 0 | 0 |
| eee. In the past 30 days, how much of your time was spent thinking about opioid medications (having enough, taking them, dosing schedule, etc.)? | 0 | 0 | 0 | 0 | 0 |
| fff. In the past 30 days, how often have you been in an argument? | 0 | 0 | 0 | 0 | 0 |
| ggg. In the past 30 days, how often have you had trouble controlling your anger (e.g., road rage, screaming, yelling, etc.)? | 0 | 0 | 0 | 0 | 0 |
| hhh. In the past 30 days, how often have you needed to take pain medications belonging to someone else? | 0 | 0 | 0 | 0 | 0 |

DATE: 6 1418 19
EXP: 6 114119
Naval Health Research Center San Diego

G-63

| iii la tha nact 20 days hayyaftan hayyay | | | | | |
|---|---|---|---|---|---|
| iii. In the past 30 days, how often have you been worried about how you're handling your medications? | 0 | 0 | 0 | 0 | 0 |
| | Never | Seldom | Sometimes | Often | Very<br>often |
| jjj. In the past 30 days, how often have others been worried about how you're handling your medications? | 0 | 0 | 0 | 0 | 0 |
| kkk. In the past 30 days, how often have<br>you had to make an emergency phone<br>call or show up at the clinic without an<br>appointment? | 0 | 0 | 0 | 0 | 0 |
| III. In the past 30 days, how often have you gotten angry with people? | 0 | 0 | 0 | 0 | 0 |
| mmm. In the past 30 days, how often have you had to take more of your medication than prescribed? | 0 | 0 | 0 | 0 | 0 |
| nnn. In the past 30 days, how often have you borrowed pain medication from someone else? | 0 | 0 | 0 | 0 | 0 |
| ooo. In the past 30 days, how often have you used your pain medicine for symptoms other than for pain (e.g., to help you sleep, improve your mood, or relieve stress)? | 0 | 0 | 0 | 0 | 0 |
| ppp. In the past 30 days, how often have you had to visit the Emergency Room? | 0 | 0 | 0 | 0 | 0 |

### HOUSEHOLD

#### 4. Please answer the following.

| Turk Summer | 9 | No | Yes |
|---|---|---|---|
| j. | Do you live with others? | 0 | 0 |
| k. | Some types of medication pose a greater risk of misuse. These include some pain medications, benzodiazepines muscle relaxants, sleeping medications, and some anxiety medications among others. Is someone in your household or living quarters taking these types of medications? | 0 | 0 |
| l. | Have you shared your prescription medication with others? | 0 | 0 |

APPROVED

DATE: 6 1 4 1 18

EXP: 6 1/4 1 19

Naval Health Research Centler San Diego

G-64

| | COMMUNI | CATION | | | |
|---|---|---|---|---|---|
| <ol><li>If you wanted to, how <u>prepared</u> do<br/>you feel to talk to?</li></ol> | Very<br>unprepared | Somewhat unprepared | Neutral | Somewhat prepared | Very<br>prepared |
| m. Someone in your chain of command if you were concerned about YOUR possible misuse of a prescribed medication? | 0 | 0 | 0 | 0 | 0 |
| n. Your <u>doctor</u> if you were concerned<br>about <u>YOUR</u> possible misuse of a<br>prescribed medication? | 0 | 0 | 0 | 0 | 0 |
| o. A <u>buddy</u> (fellow service member) if you were concerned about <u>THEIR</u> possible misuse of a prescribed medication? | 0 | 0 | 0 | 0 | 0 |
| p. A <u>spouse</u> (or significant other) if you were concerned about <u>THEIR</u> possible misuse of a prescribed medication? | 0 | 0 | 0 | 0 | 0 |

#### **ATTITUDES**

# 6. Please indicate how much you agree or disagree with the statements.

| | Strongly<br>disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Strongly<br>agree |
|---|---|---|---|---|---|
| ooo. Misusing prescription drugs is dangerous. | 0 | 0 | 0 | 0 | 0 |
| ppp. Most service members misuse<br>prescription drugs at some point while<br>active duty. | on O | 0 | 0 | 0 | 0 |
| qqq. It's not a big deal to share prescript medication with someone if you're tryi to help them. | | 0 | 0 | 0 | 0 |
| rrr. It should be illegal to share prescription medication with friends. | 0 | 0 | 0 | 0 | 0 |
| sss.lt should be illegal to share prescription medication with family members. | 0 | 0 | 0 | 0 | 0 |
| ttt. If you've been prescribed medication be your doctor, you should take it only as directed. | y ○ | 0 | O APPRO DATE: 6 / 4 EXP: 6 //4 | 0<br>1/8<br>1/8 JLI | |
| N D LANANZONO | G-03 | L | Naval Health Research | h Center San Diego | |

| | | | трр, т тотооо | | |
|---|---|---|---|---|---|
| uuu. If you share your prescription medications with friends or family, you are putting their health at risk. | 0 | 0 | 0 | 0 | 0 |
| | Strongly<br>disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Strongly<br>agree |
| vvv. The risk of getting in trouble for taking pain medication differently than prescribed is a concern for me. | 0 | 0 | 0 | 0 | 0 |
| www. There is a high risk of getting caught if you take your own old prescription medication. | 0 | 0 | 0 | 0 | 0 |
| xxx. Using someone else's prescription medication can be hazardous to your health. | 0 | 0 | 0 | 0 | 0 |
| yyy. Using someone else's prescription medication can cost you your military career. | 0 | 0 | 0 | 0 | 0 |
| zzz.It is no big deal if I take a higher dose of<br>my prescription pain reliever than<br>directed. | 0 | 0 | 0 | 0 | 0 |
| aaaa. It is risky to my health to take my medication more often than prescribed. | 0 | 0 | 0 | 0 | 0 |
| bbbb. Even if a medication label says not to<br>take it with alcohol, it is ok to take it with<br>only one drink. | 0 | 0 | 0 | 0 | 0 |
| cccc. Drinking alcohol with prescription pain relievers is only risky if you are binge drinking. | 0 | 0 | 0 | 0 | 0 |
| dddd. If I have questions about a prescription medication, I should ask my provider. | 0 | 0 | 0 | 0 | 0 |
| eeee. If I have questions about a prescription medication, I should ask the pharmacy tech. | 0 | 0 | 0 | 0 | 0 |
| ffff. It is important to read the label on my prescription medication. | 0 | 0 | 0 | 0 | 0 |
| gggg. It is important to read the material that the pharmacy provides with my prescription medication. | 0 | 0 | 0 | 0 | 0 |
| hhhh. If I have concerns about my medication, it's important that I know where to go for information. | 0 | 0 | 0 | 0 | 0 |
| iiii. It is ok to use your leftover prescription medication for a new condition. | 0 | 0 | 0 | 0 | 0 |
| jjjj. There is nothing wrong with taking an<br>extra dose of my prescription pain reliever<br>if I am in pain. | 0 | ° | DATE: 6 14 | 0<br>VED<br>1/8 | |
| Version Date: 14 MAY 2019 | G-66 | | EXP: 6 1/4 Naval Health Research | 1 19<br>h Center San Diego | , |

# 7. Please indicate how much you agree or disagree with the statements.

| | Strongly<br>disagree | Disagree | Neither agree nor disagree | Agree | Strongly<br>agree |
|---|---|---|---|---|---|
| y. There are certain situations where it is ok to take someone else's prescribed medication. | 0 | 0 | 0 | 0 | 0 |
| If a person is in physical pain from an injury, taking someone else's prescription medication is okay. | 0 | 0 | 0 | 0 | 0 |
| aa. As long as it makes you feel better and not<br>worse, it's fine to take prescription drugs<br>while drinking. | 0 | 0 | 0 | 0 | 0 |
| bb. An individual should only take medication<br>that is prescribed to them by a medical<br>professional. | 0 | 0 | 0 | 0 | 0 |
| cc. It is acceptable for a fellow service member to borrow someone's prescription medication in order to enhance their readiness. | 0 | 0 | 0 | 0 | 0 |
| dd. It is ok for a service member to take medication that is not prescribed to them in order to decrease appetite and lose weight. | 0 | 0 | 0 | 0 | 0 |
| ee. Using prescribed medications to stay awake for duty is okay. | 0 | 0 | 0 | 0 | 0 |
| ff. Taking medication that is not prescribed to<br>you should be illegal. | 0 | 0 | 0 | 0 | 0 |

## 8. How much do you think people <u>risk harming themselves</u> (physically or in other ways) by...?

| | No risk | Slight risk | Moderate<br>risk | Great risk |
|---|---|---|---|---|
| p. Taking <u>someone else's</u> prescription drug (examples: oxycodone, Valium)? | 0 | O | OPROVED | 0 |
| G-67 | | DATE: 6 EXP: 6 Naval Health Ro | 141/8<br>1/41/9<br>search Center San I | n D<br>Diego |

| Hurtado, Evaluation of a Di | ug Abuse Educ | ational App, Pro | tocol # NHRC | .2016.0019 |
|---|---|---|---|---|
| q. Taking a prescription drug (examples: oxycodone,<br>Valium) in <u>higher doses</u> than what a doctor<br>prescribed? | 0 | 0 | 0 | 0 |
| r. Taking a prescription drug (examples: oxycodone, Valium) together with alcohol or other drugs? | 0 | 0 . | 0 | 0 |
| s. Having 5 or more drinks of alcohol once or twice each weekend? | 0 | 0 | 0 | 0 |
| t. Smoking marijuana regularly (more than once a | 0 | 0 | 0 | 0 |
| week)? | | | | |
| week)? 9. Please indicate how much you agree or disagree | with the stat | ements. | | |
| | with the stat<br>Strongly<br>disagree | ements.<br>Disagree | Agree | Strongly<br>agree |
| | Strongly | | Agree<br>O | ٠. |
| <ul> <li>9. Please indicate how much you agree or disagree</li> <li>m. I have made a final decision to stay away from misusing prescription drugs (examples:</li> </ul> | Strongly<br>disagree | Disagree | | agree |

#### KNOWLEDGE

0

0

10.Based upon DoD policy, which of the following is **NOT** an example of prescription drug misuse?

p. Taking more of your medication that is prescribed

exactly as prescribed by my provider.

prescription medication.

p. I plan to intervene if I see someone misusing

q. Taking your medication at 2150 instead of 2200 because you plan to go to sleep

r. Using the prescription you got earlier this year for your knee for a back strain you got this week

s. Taking your pain medication 4 times a day instead of 3 like it says on the label

t. Giving some of your medication to your spouse because he or she ran out

**11.** Which of the following is <u>NOT</u> a recommendation in the Prescription for Discharge campaign to protect Sailors and Marines from prescription drug misuse/abuse?

p.Report promptly

q. Take correctly

r. Save for emergencies

s. Never share

APPROVED

DATE: 6 14 118 775

EXP: 6 114 1 19

Naval Health Research Center San Diego

0

0

G-68

- t. Dispose properly
- **12.** What should a service member do if they receive a prescription medication from a *non-military* medical treatment facility?
- p.Report it to the Chaplain
- q.It ONLY needs to be reported to their military health care provider if they had an adverse reaction
- r. It does not need to be reported
- s. Report it to their military health care provider at their next visit
- t. Report it to their chain of command and ensure it is entered into their military health record
- 13. What type of alternative treatment involves visualizing specific positive scenes to reduce stress?
- p.Biofeedback
- q.Acupuncture
- r. Yoga
- s. Guided Imagery
- t. Physical Therapy
- 14. What type of alternative treatment involves becoming mindful of one's thoughts and sensations in a nonjudgmental way?
- p. Physical Therapy
- q.Biofeedback
- r. Chiropractic Therapies
- s. Massage Therapy
- t. Meditation
- **15.** What can you do if you suspect someone is misusing prescription medication?
- p. Provide support
- q.Be a role model
- r. Keep medications safe and secured
- s. Inform chain of command or law enforcement officials
- t. All of the above
- 16. Which of the following is NOT potentially a sign or symptom associated with prescription drug misuse?
  - p.Relationship problems
  - q.Sudden weight loss or gain
  - r. Asking your doctor questions about your prescription
  - s. Changes in appetite or sleep patterns
  - t. Decreased performance at work
- 17. What are the two most commonly misused prescription drugs among military personnel?
  - m. Pain relievers (opioids) and central nervous system depressants (sedatives)
  - n. Pain relievers (opioids) and protease inhibitors
  - o.Central nervous system depressants (sedatives) and protease inhibitors
  - p.Central nervous system depressants (sedatives) and central nervous system stimulants
    Pain relievers (opioids) and central nervous system stimulants
- 18. Which of the following is a negative consequence of misusing prescription drugs?
  - p.Drug addiction
  - q.Altered judgment

APPROVED

DATE: 6 14 1/8

EXP: 6 1/41/9

Naval Health Research Center San Diego

G-69

- r. Unintentional overdose
- s. Drug tolerance
- t. All of the above
- **19.** What is a specific sign or symptom of prescription drug misuse?
  - p. Faking illness or injury to obtain medications
  - q. Excessive visits to the doctor
  - r. Stealing, forging, or selling prescriptions
  - s. None of the above
  - t. All of the above

DATE: 6 14 118 TU

EXP: 6 114 19

Naval Health Research Center San Diego

- 20. Which of the following could help you reduce your risk of prescription drug misuse? (Select the best answer)
  - p. Ask your friend which medication worked best for them to treat pain
  - q. Take your old prescription for pain without consulting your doctor
  - r. Wait until your pain is unbearable before taking pain medication instead of taking it at the regular intervals indicated
  - s. Talk to your doctor about symptoms you may be having or concerns about your medication
  - t. Mix your prescription medication with over-the-counter medicine and supplements
- 21. It is important to talk to your doctor or pharmacist about... (Select the best answer)
  - p. Using over-the-counter medications while using your prescription
  - q.Supplements that you routinely take
  - r. Symptoms and side effects you are experiencing
  - s. A and C
  - t. All of the above
- 22. TRUE OR FALSE: Everyday activities such as playing sports cannot cause traumatic brain injuries (TBI).
  - g.TRUE
  - h.FALSE
- 23. TRUE OR FALSE: Prescription drugs are regulated so they are always safe to take.
  - g.TRUE
  - h.FALSE
- 24. TRUE OR FALSE: It is safe to take prescription medication from a previous health problem to treat new symptoms.
  - g. TRUE
  - h.FALSE
- 25. Which of the following is a good resource for someone seeking information about a prescription medication misuse problem? (Select all that apply)
- p.SACO or DAPA
- q.Corpsman or other medical provider
- r. Commanding Officer
- s. Diversity Officer
- t. MilitaryOneSource
- 26. Drinking alcohol with prescription medication can do which of the following? (Select all that apply)
  - p.Increase side effects
  - q.Increase effectiveness
  - r. Decrease effectiveness
  - s. Decrease sedative effects
  - t. Increase risk of a toxic reaction

APPROVED

DATE: 6 14 1/8

EXP: 6 1/4 1/9

Naval Health Research Center San Diego

- 27. Which of the following has contributed to the increase in prescription drug abuse among service members? (Select all that apply)
  - p.Increase in prescriptions for pain related to injuries among OIF and OEF veterans
  - q.Decrease in military pharmacy regulations
  - r. Increase in average working hours among service members
  - s. Decrease in the number of compounds tested in drug screening
  - t. Increase in the number of military health care providers
- 28. Which step(s) can you take to reduce prescription drug misuse? (Select all that apply)
  - p. Use previously prescribed medication for a current health issue
  - q. Keep your medications safe and secured
  - r. Only borrow prescription medication from a spouse or other trusted source
  - s. Dispose of unused or expired prescription medication properly
  - t. Do not share medication
- 29. Which of the following are key points you would want to discuss with your pharmacist when getting a new prescription? (Select all that apply)
  - p. Best time of day to take medication
  - q.Other health conditions the medication may be used for in the future
  - r. Prescribed dosage
  - s. Potential side effects and warnings
  - t. Alternative non-medical treatments
- 30. Which of the following are signs and symptoms of depression? (Select all that apply)
  - p.Changes in appetite or weight
  - q.Increased motivation
  - r. Increased energy
  - s. Decreased energy
  - t. Irritability
- **31.** Which of the following statement(s) about sleep is TRUE? (Select all that apply)
  - p. The quality of sleep you are getting is just as important as the amount
  - q.Sleep problems can be a side effect of some medications
  - r. The amount of sleep you are getting is the most important aspect of sleep
  - s. Sleep problems can be a symptom of a mental health condition
  - t. Catching-up on sleep is just as effective as regular sleep
- **32.**What are two common forms of treatment for mental health conditions such as depression, anxiety, and PTSD? (Select all that apply)
  - p.Medication
  - q.Physical therapy
  - r. Dietary changes
  - s. No treatment available
  - t. Psychotherapy

#### **SUBMIT SURVEY**

Thanks for completing this survey! We greatly appreciate your participation!


DATE: 6 14 118 TU